CLINICAL TRIAL: NCT01970865
Title: PHASE 1/2 STUDY OF PF-06463922 (AN ALK/ROS1 TYROSINE KINASE INHIBITOR) IN PATIENTS WITH ADVANCED NON-SMALL CELL LUNG CANCER HARBORING SPECIFIC MOLECULAR ALTERATIONS
Brief Title: A Study Of PF-06463922 An ALK/ROS1 Inhibitor In Patients With Advanced Non Small Cell Lung Cancer With Specific Molecular Alterations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7461001; 2013-002620-17 (EudraCT Number)
Expanded Access: NCT03127618 (Approved for marketing)
Record Dates: First submitted 2013-10-16; First posted 2013-10-28 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: ALK-positive Non Small Cell Lung Cancer (NSCLC) and ROS1-positive NSCLC
Keywords: Phase 1; Phase 2; safety; pharmacokinetic; pharmacodynamic; efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06463922 (Experimental)
  Interventions: Drug: PF-06463922
- Crizotinib (Other): ALK+ NSCLC patients who are treatment naïve may be eligible to receive crizotinib following PF-06463922 as a substudy to the main study.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: PF-06463922 — Oral, starting dose 10mg once a day, dose escalation in Phase 1 until recommended Phase 2 dose determined, continuous daily dosing, cycles lasting 21 days
  Arms: PF-06463922
Drug: Crizotinib — Oral, starting dose of 250 mg BID continuous daily dosing every 21 days
  Other Names: Xalkori
  Arms: Crizotinib

SUMMARY:
Phase 1 and 2 trial to study the safety, pharmacokinetics, pharmacodynamics, patient reported outcomes and efficacy of PF-06463922 in ALK + advanced non-small cell lung cancer patients and ROS1+ advanced non small cell lung cancer patients .

ELIGIBILITY:
Inclusion Criteria

* Evidence of histologically or cytologically confirmed diagnosis of metastatic NSCLC (Stage IV, AJCC v7.0) that carries an ALK rearrangement, as determined by the Food and Drug Administration (FDA) approved FISH assay (Abbott Molecular Inc) or by Immunohistochemistry (IHC) (Ventana Inc), or a ROS1 rearrangement as determined by FISH or RT PCR or Next Generation Sequencing (NGS) via a local diagnostic test (LDT). All patients (ALK positive and ROS1 positive) must have archival tissue sample available and collected prior to enrollment.
* Disease Status Requirements:

Phase 1: ALK-positive NSCLC and ROS1-positive patients must either be treatment naïve in the advanced setting or have had disease progression after at least 1 previous ALK/ROS1 inhibitor therapy(ies).

Phase 2:

ALK-positive NSCLC patients must either be or have had:

* Treatment naïve (ie, no prior chemotherapy in the metastatic disease setting and no prior ALK inhibitor therapy allowed).
* Disease progression after crizotinib only. No prior chemotherapy is allowed in the metastatic disease setting.
* Disease progression after crizotinib and 1 or 2 prior regimens of chemotherapy in the metastatic disease setting.
* Disease progression after 1 prior ALK inhibitor therapy other than crizotinib. Patients may have had any number of prior chemotherapy regimens in any disease setting.
* Disease progression after 2 prior ALK inhibitor therapies. Patients may have had any number of prior chemotherapy regimens in any disease setting.
* Disease progression after 3 prior ALK inhibitor therapies. Patients may have had any number of prior chemotherapy regimens in any disease setting.

ROS1-positive NSCLC patients may be:

* Treatment naïve (ie, no prior chemotherapy in the metastatic disease setting and no prior ROS inhibitor therapy).
* Any number of prior therapies (ie, chemotherapy and/or ROS inhibitor therapies).

  * Tumor Requirements:

All Patients must have at least one measurable target extracranial lesion according to RECIST v1.1. In addition patients with asymptomatic CNS metastases (including patients asymptomatic by means of stable or decreasing doses of steroids within the last 2 weeks prior to study entry) will be eligible. Patients who have leptomeningeal disease (LM) or carcinomatous meningitis (CM) are eligible.

* Adequate Bone Marrow, Pancreatic Function, Renal Function and Liver Function.
* Negative Serum pregnancy test for females of childbearing potential Exclusion Criteria
* Radiation therapy (except palliative to relieve bone pain) within 2 weeks of study entry. Whole brain radiation must have completed at least 4 weeks prior to study entry.
* Systemic anti cancer therapy completed within a minimum of 5 half lives of study entry.
* Prior therapy with an antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including, but not limited to, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T lymphocyte associated antigen 4 (anti-CTLA-4) antibody.
* Active and clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) related illness.
* Clinically significant cardiovascular disease (that is, active or <3 months prior to enrollment): cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec. Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, etc.), machine-read ECG with QTc >470 msec, or congenital long QT syndrome.
* History of extensive, disseminated, bilateral or presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis.
* Current use or anticipated need for food or drugs that are known strong or moderate CYP3A4 inhibitors, inducers and substrates; drugs that are CYP2C9 substrates; drugs that are sensitive CYP2B6 substrates; drugs that are strong CYP2C19 inhibitors; drugs that are strong CYP2C8 inhibitors; and drugs that are P-gp substrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (73):
- United States (30):
  - Highlands Oncology Group/Research, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Chao Family Comprehensive Cancer Center, Orange, California
  - UC Irvine Medical Center, Orange, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavillion (AOP), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - MDZ: Yale-New Haven Hospital, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Center Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Siteman Cancer Center-West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Rockefeller Patient Pavilion - Memorial Sloan Kettering, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Rochester Regional Health System, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - The Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute (Pharmacy), Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Australia (5):
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney Local Health District [rpa], New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- University Hospital Antwerp, Edegem, Belgium
- Canada (3):
  - British Columbia Cancer Agency-Vancouver Centre, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (6):
  - CHU Grenoble/ Hôpital Albert Michallon, Grenoble
  - CHU de Rennes - Hôpital Pontchaillou - CIC Inserm, Rennes
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Institut Universitaire du Cancer de Toulouse (IUCT-O), Toulouse
  - Institut Gustave Roussy (comite poumon-pneumologie), Villejuif
  - Institut Gustave Roussy- Pharmacie-Unite Essais Cliniques, Villejuif
- Universitaetsklinik Koeln, Cologne, Germany
- Department of Clinical Oncology, Prince of Wales Hospital, Shatin, Hong Kong
- Italy (4):
  - Struttura Operativa Complessa Oncologia, Aviano (PN)
  - Dipartimento di Oncologia Medica, UO Medicina 1Q A, Unita' Nuovi Farmaci e Terapie Innovative, Milan
  - Unita di Farmacologia Clinica e Nuovi Farmaci, Milan
  - Oncologia Medica, Perugia
- Japan (11):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kindai University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- Singapore (3):
  - National University Hospital, Singapore
  - National University Hospital Medical Centre, Singapore
  - National Cancer Center, Singapore
- Seoul National University Hospital / Department of Internal Medicine, Seoul, South Korea
- Spain (4):
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad De Navarra, Pamplona, Navarre
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital Universitari de la Vall D'Hebron Edificio General. Planta Baja. UITM. Servicio de Oncologia, Barcelona
- Switzerland (2):
  - Hospital of Lausanne (CHUV), Lausanne
  - Kantonsspital Winterthur, Winterthur
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ou SI, Solomon BJ, Besse B, Bearz A, Lin CC, Chiari R, Camidge DR, Lin JJ, Abbattista A, Toffalorio F, Soo RA. Final Overall Survival and Long-Term Safety of Lorlatinib in Patients With ALK-Positive NSCLC From the Pivotal Phase 2 Study: A Brief Report. J Thorac Oncol. 2025 Apr;20(4):513-520. doi: 10.1016/j.jtho.2024.11.021. Epub 2024 Nov 22. PMID 39581380
- [Derived] Chen J, Bearz A, Kim DW, Mamdani H, Bauman J, Chiari R, Ou SI, Solomon BJ, Soo RA, Felip E, Shaw AT, Thurm H, Clancy JS, Lee K, O'Gorman M, Tanski C, Pithavala YK. Evaluation of the Effect of Lorlatinib on CYP2B6, CYP2C9, UGT, and P-Glycoprotein Substrates in Patients with Advanced Non-Small Cell Lung Cancer. Clin Pharmacokinet. 2024 Feb;63(2):171-182. doi: 10.1007/s40262-023-01309-4. Epub 2023 Dec 11. PMID 38079095
- [Derived] Dagogo-Jack I, Abbattista A, Murphy JF, Krulewicz S, Do A, Peterson J, Lin JJ, Gainor JF, Messina R, Krueger EA, Thurm H, Yeap BY. Factors Associated With Developing Neurocognitive Adverse Events in Patients Receiving Lorlatinib After Progression on Other Targeted Therapies. J Thorac Oncol. 2023 Jan;18(1):67-78. doi: 10.1016/j.jtho.2022.09.219. Epub 2022 Sep 29. PMID 36184067
- [Derived] Soo RA, Huat Tan E, Hayashi H, Seto T, Lin CC, Ou SI, Kim DW, Liu G, Abbattista A, Martini JF, Hooi Wong C, Toffalorio F, Solomon BJ. Efficacy and safety of lorlatinib in Asian and non-Asian patients with ALK-positive advanced non-small cell lung cancer: Subgroup analysis of a global phase 2 trial. Lung Cancer. 2022 Jul;169:67-76. doi: 10.1016/j.lungcan.2022.05.012. Epub 2022 May 23. PMID 35660971
- [Derived] Ou SI, Solomon BJ, Shaw AT, Gadgeel SM, Besse B, Soo RA, Abbattista A, Toffalorio F, Wiltshire R, Bearz A. Continuation of Lorlatinib in ALK-Positive NSCLC Beyond Progressive Disease. J Thorac Oncol. 2022 Apr;17(4):568-577. doi: 10.1016/j.jtho.2021.12.011. Epub 2022 Jan 10. PMID 35026476
- [Derived] Chen J, Ruiz-Garcia A, James LP, Peltz G, Thurm H, Clancy J, Hibma J. Lorlatinib Exposure-Response Analyses for Safety and Efficacy in a Phase I/II Trial to Support Benefit-Risk Assessment in Non-Small Cell Lung Cancer. Clin Pharmacol Ther. 2021 Nov;110(5):1273-1281. doi: 10.1002/cpt.2228. Epub 2021 Jun 26. PMID 33973232
- [Derived] Chen J, O'Gorman MT, James LP, Klamerus KJ, Mugundu G, Pithavala YK. Pharmacokinetics of Lorlatinib After Single and Multiple Dosing in Patients with Anaplastic Lymphoma Kinase (ALK)-Positive Non-Small Cell Lung Cancer: Results from a Global Phase I/II Study. Clin Pharmacokinet. 2021 Oct;60(10):1313-1324. doi: 10.1007/s40262-021-01015-z. Epub 2021 May 3. PMID 33937954
- [Derived] Peters S, Shaw AT, Besse B, Felip E, Solomon BJ, Soo RA, Bearz A, Gadgeel SM, Lin CC, Kao S, Seto T, Masters ET, Abbattista A, Clancy JS, Thurm H, Reisman A, Peltz G, Ross Camidge D. Impact of lorlatinib on patient-reported outcomes in patients with advanced ALK-positive or ROS1-positive non-small cell lung cancer. Lung Cancer. 2020 Jun;144:10-19. doi: 10.1016/j.lungcan.2020.02.011. Epub 2020 Mar 10. PMID 32344248
- [Derived] Bauer TM, Shaw AT, Johnson ML, Navarro A, Gainor JF, Thurm H, Pithavala YK, Abbattista A, Peltz G, Felip E. Brain Penetration of Lorlatinib: Cumulative Incidences of CNS and Non-CNS Progression with Lorlatinib in Patients with Previously Treated ALK-Positive Non-Small-Cell Lung Cancer. Target Oncol. 2020 Feb;15(1):55-65. doi: 10.1007/s11523-020-00702-4. PMID 32060867
- [Derived] Shaw AT, Solomon BJ, Chiari R, Riely GJ, Besse B, Soo RA, Kao S, Lin CC, Bauer TM, Clancy JS, Thurm H, Martini JF, Peltz G, Abbattista A, Li S, Ou SI. Lorlatinib in advanced ROS1-positive non-small-cell lung cancer: a multicentre, open-label, single-arm, phase 1-2 trial. Lancet Oncol. 2019 Dec;20(12):1691-1701. doi: 10.1016/S1470-2045(19)30655-2. Epub 2019 Oct 25. PMID 31669155
- [Derived] Solomon BJ, Besse B, Bauer TM, Felip E, Soo RA, Camidge DR, Chiari R, Bearz A, Lin CC, Gadgeel SM, Riely GJ, Tan EH, Seto T, James LP, Clancy JS, Abbattista A, Martini JF, Chen J, Peltz G, Thurm H, Ou SI, Shaw AT. Lorlatinib in patients with ALK-positive non-small-cell lung cancer: results from a global phase 2 study. Lancet Oncol. 2018 Dec;19(12):1654-1667. doi: 10.1016/S1470-2045(18)30649-1. Epub 2018 Nov 6. PMID 30413378
- [Derived] Shaw AT, Felip E, Bauer TM, Besse B, Navarro A, Postel-Vinay S, Gainor JF, Johnson M, Dietrich J, James LP, Clancy JS, Chen J, Martini JF, Abbattista A, Solomon BJ. Lorlatinib in non-small-cell lung cancer with ALK or ROS1 rearrangement: an international, multicentre, open-label, single-arm first-in-man phase 1 trial. Lancet Oncol. 2017 Dec;18(12):1590-1599. doi: 10.1016/S1470-2045(17)30680-0. Epub 2017 Oct 23. PMID 29074098
- [Derived] Shaw AT, Friboulet L, Leshchiner I, Gainor JF, Bergqvist S, Brooun A, Burke BJ, Deng YL, Liu W, Dardaei L, Frias RL, Schultz KR, Logan J, James LP, Smeal T, Timofeevski S, Katayama R, Iafrate AJ, Le L, McTigue M, Getz G, Johnson TW, Engelman JA. Resensitization to Crizotinib by the Lorlatinib ALK Resistance Mutation L1198F. N Engl J Med. 2016 Jan 7;374(1):54-61. doi: 10.1056/NEJMoa1508887. Epub 2015 Dec 23. PMID 26698910
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7461001&StudyName=A%20Study%20Of%20PF-06463922%20An%20ALK/ROS1%20Inhibitor%20In%20Patients%20With%20Advanced%20Non%20Small%20Cell%20Lung%20Cancer%20With%20Specific%20Molecular%20Alterations

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 364 participants were enrolled in this study.
Groups:
- 10 mg QD (Phase 1): PF-06463922 10 mg was orally given once daily (QD) on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 25 mg QD (Phase 1): PF-06463922 25 mg was orally given QD in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal. Midazolam 2 mg was orally given QD on Day -7 and Cycle 1 Day 15.
- 50 mg QD (Phase 1): PF-06463922 50 mg was orally given QD on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 75 mg QD (Phase 1): PF-06463922 75 mg was orally given QD on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 100 mg QD (Phase 1): PF-06463922 100 mg was orally given QD on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 150 mg QD (Phase 1): PF-06463922 150 mg was orally given QD in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal. Midazolam 2 mg was orally given QD on Day -7 and Cycle 1 Day 15.
- 200 mg QD (Phase 1): PF-06463922 200 mg was orally given QD on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 35 mg BID (Phase 1): PF-06463922 35 mg was orally given twice daily (BID) on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 75 mg BID (Phase 1): PF-06463922 75 mg was orally given BID on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- 100 mg BID (Phase 1): PF-06463922 100 mg was orally given BID on Day -7 and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-1 (Phase 2): Treatment-naïve participants with advanced anaplastic lymphoma kinase (ALK)-positive non-small-cell lung cancer (NSCLC) with or without asymptomatic central nervous system (CNS) metastases were given PF-06463922 100 mg orally QD on Day -7 (only participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-2 (Phase 2): Participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after only crizotinib therapy were given PF-06463922 100 mg orally QD on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-3 (Phase 2): Participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after crizotinib therapy and 1 or 2 prior regimens of chemotherapy given before or after crizotinib therapy, or participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after 1 ALK inhibitor therapy other than crizotinib with or without any number of prior chemotherapy regimens in any disease setting were given PF-06463922 100 mg orally QD on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-4 (Phase 2): Participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after 2 prior lines of ALK inhibitor therapies were given PF-06463922 100 mg orally QD on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-5 (Phase 2): Participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after 3 prior lines of ALK inhibitor therapies were given PF-06463922 100 mg orally QD on Day -7 (only for participant scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-6 (Phase 2): Participants with advanced ROS1-positive NSCLC who were treatment naïve or had any number of prior cancer therapies with or without asymptomatic CNS metastases were given PF-06463922 100 mg orally QD on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- Japan Lead-In Cohort (LIC): Few Japanese participants were given PF-06463922 100 mg orally once daily (QD) in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal to evaluate safety of PF-06463922 in Japanese participants, in order to support inclusion of Japanese participants in Phase 2.
- Drug-drug Interaction (DDI) Sub-study: Participants with advanced ALK positive or ROS1-positive NSCLC who were treatment naïve or had any number of prior cancer therapies with or without asymptomatic CNS metastases were administered a single dose of a probe substrate alone on Day -2. Participants were given PF-06463922 100 mg orally QD starting on Cycle1 Day 1 and along with probe substrate on Day 15 Cycle 1.
Period: Overall Study
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | Japan Lead-In Cohort (LIC) | Drug-drug Interaction (DDI) Sub-study
Started | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 65 | 46 | 47 | 3 | 32
Completed | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 2 | 18 | 7 | 18 | 8 | 3 | 7 | 2 | 6
Not Completed | 3 | 3 | 3 | 10 | 14 | 3 | 3 | 3 | 2 | 2 | 12 | 20 | 42 | 57 | 43 | 40 | 1 | 26
Not completed — Death | 3 | 2 | 3 | 6 | 9 | 3 | 2 | 3 | 2 | 2 | 8 | 13 | 25 | 46 | 37 | 22 | 1 | 17
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 4 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 8 | 3 | 2 | 3 | 0 | 2
Not completed — Participant refused further follow-up | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 7 | 8 | 3 | 11 | 0 | 6

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled patients who receive at least one dose of PF-06463922 (including Lead-in dose).
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | Japan Lead-In Cohort (LIC) | Drug-drug Interaction (DDI) Sub-study | Total
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 65 | 46 | 47 | 3 | 32 | 364
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 0 | 1 | 0 | 5 | 7 | 1 | 1 | 0 | 0 | 2 | 4 | 5 | 14 | 19 | 13 | 12 | 2 | 5 | 91
  45-64 years | 1 | 1 | 3 | 6 | 9 | 1 | 2 | 2 | 2 | 1 | 18 | 13 | 34 | 37 | 26 | 27 | 1 | 20 | 204
  >=65 years | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 8 | 9 | 12 | 9 | 7 | 8 | 0 | 7 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 7 | 11 | 2 | 2 | 2 | 3 | 2 | 13 | 17 | 38 | 37 | 25 | 27 | 2 | 15 | 206
  Male | 1 | 3 | 2 | 5 | 6 | 1 | 1 | 1 | 0 | 2 | 17 | 10 | 22 | 28 | 21 | 20 | 1 | 17 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 2 | 2 | 3 | 7 | 13 | 2 | 2 | 1 | 2 | 3 | 10 | 13 | 25 | 32 | 27 | 25 | 0 | 21 | 190
  BLACK | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 6
  ASIAN | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 17 | 10 | 23 | 23 | 14 | 16 | 3 | 11 | 124
  Others | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 2 | 3 | 0 | 0 | 13
  Unspecified | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 10 | 7 | 3 | 2 | 0 | 0 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cycle 1 Dose-Limiting Toxicities (DLTs) in Phase 1
Description: DLT: any of following adverse events (AEs) attributable to PF-06463922: (1) hematologic: grade 4 neutropenia for >7 days; febrile neutropenia; grade>=3 neutropenic infection; grade>=3 thrombocytopenia with bleeding; grade 4 thrombocytopenia; (2) non-hematologic: grade>=3 pancreatitis; grade>=3 toxicities (excluding grade >=3 laboratory abnormalities not requiring dose modifications) persisting after optimal treatment with standard medical therapy; symptomatic grade >=3 QT interval corrected for heart rate (QTc) prolongation, or asymptomatic grade >=3 prolongation that had been confirmed by repeat testing, re-evaluation by qualified person, persisted after correction of reversible causes; >=20% decrease from baseline in left ventricular ejection fraction (LVEF); (3) other: failure to deliver at least 16 out of 21 prescribed daily total dose due to toxicities attributable to study drug; failure to restart dosing after 21 days (1 cycle) delay due to toxicity attributable to study drug.
Time Frame: Cycle 1 (21 days)
Population: Maximum Tolerated Dose (MTD) evaluable population included all enrolled participants who received at least 75% of the planned PF-06463922 doses in Cycle 1. Participants who received less than 75% of the planned PF-06463922 doses in Cycle 1 due to DLT were also considered evaluable for MTD. Here, "Overall Number Analyzed" signifies participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 3 | 11 | 16 | 3 | 3 | 2 | 3 | 3
Participants
  With DLT | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  No DLT | 3 | 2 | 3 | 6 | 8 | 2 | 1 | 2 | 3 | 2
  Data missing | 0 | 1 | 0 | 5 | 8 | 1 | 1 | 0 | 0 | 1

2. Primary Outcome: Percentage of Participants With Overall and Intracranial Objective Response (Phase 2)
Description: Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. Intracranial OR refers to confirmed CR or PR considering only lesions within brain. CR was defined as the disappearance of all non-lymph node target lesions (where all target lesions are recorded with a length of 0 milliliter (mm) on Target Lesions electronic case report form (eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as a 30 percent (%) or more decrease in sum of lesion dimensions (SLD) of target lesions, taking as reference the baseline SLD. Results presented here were based on independent central review.
Time Frame: 3 years
Population: The intent-to-treat (ITT) analysis set was used for overall response assessment, and included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922; participants with central nervous system (CNS) metastases in the ITT analysis set were used for intracranial response assessment. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 30 | 27 | 60 | 65 | 46 | 47
Percentage of participants
  Objective response: number analyzed (Participants) | 30 | 27 | 59 | 65 | 46 | 47
  Objective response | 90.0 [73.5 to 97.9] | 74.1 [53.7 to 88.9] | 50.8 [37.5 to 64.1] | 41.5 [29.4 to 54.4] | 34.8 [21.4 to 50.2] | 36.2 [22.7 to 51.5]
  Intracranial objective response: number analyzed (Participants) | 8 | 17 | 32 | 45 | 38 | 25
  Intracranial objective response | 75.0 [34.9 to 96.8] | 58.8 [32.9 to 81.6] | 62.5 [43.7 to 78.9] | 55.6 [40.0 to 70.4] | 39.5 [24.0 to 56.6] | 56.0 [34.9 to 75.6]

3. Secondary Outcome: Percentage of Participants With Overall and Intracranial Objective Response (Phase 1)
Description: Objective response (OR) refers to confirmed CR or PR according to RECIST version 1.1. Intracranial OR refers to confirmed CR or PR considering only lesions within brain. CR was defined as the disappearance of all non-lymph node target lesions (where all target lesions are recorded with a length of 0 mm on Target Lesions eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as a 30 % or more decrease in SLD of target lesions, taking as reference the baseline SLD. Results presented here were based on independent central review.
Time Frame: From start of study treatment until CR or PR (maximum of 8 years approximately)
Population: The ITT analysis set was used for overall response assessment and included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922; participants with CNS metastases in the ITT analysis set was used for intracranial response assessment. Here, "Number Analyzed" signifies participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- ALK Positive Population (Phase 1): This reporting arm includes all Phase 1 participants who had documented ALK rearrangement.
- ROS1 Positive Population (Phase 1): This reporting arm includes all Phase 1 participants who had documented ROS1 rearrangement.
Arm/Group | ALK Positive Population (Phase 1) | ROS1 Positive Population (Phase 1)
Number analyzed (Participants) | 41 | 12
Percentage of participants
  Objective response | 39.0 [24.2 to 55.5] | 50.0 [21.1 to 78.9]
  Intracranial objective response: number analyzed (Participants) | 34 | 8
  Intracranial objective response | 41.2 [24.6 to 59.3] | 50.0 [15.7 to 84.3]

4. Secondary Outcome: Time to Tumor Response (TTR) and Intracranial TTR (Phase 1)
Description: Time to tumor response (TTR) was defined as the time from the first dose of study treatment to the first documentation of objective tumor response (CR or PR). For participants whose objective response proceeded from PR to CR, the onset of PR was taken as the onset of response. CR was defined as the disappearance of all non-lymph node target lesions (where all target lesions are recorded with a length of 0 mm on Target Lesions eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as a 30 % or more decrease in SLD of target lesions, taking as reference the baseline SLD. TTR was only calculated for the subgroup of participants with a confirmed objective tumor response. Intracranial TTR was only calculated for participants with confirmed intracranial objective response. Results presented here were based on independent central review.
Time Frame: From start of study treatment to the first documentation of objective tumor response (CR or PR) (maximum of 8 years approximately)
Population: TTR analysis set included all ITT participants who had confirmed objective response; intracranial TTR analysis set included all ITT participants who had CNS metastases and achieved confirmed intracranial objective response.
Measure: Median (Full Range); unit: Months
Arm/Group | ALK Positive Population (Phase 1) | ROS1 Positive Population (Phase 1)
Number analyzed (Participants) | 16 | 6
Months
  TTR | 1.4 [1.2 to 15.2] | 1.4 [1.2 to 2.8]
  Intracranial TTR: number analyzed (Participants) | 14 | 4
  Intracranial TTR | 1.4 [1.2 to 20.1] | 1.4 [1.1 to 2.8]

5. Secondary Outcome: Number of Participants With Duration of Response (DOR) and Intracranial DOR (Phase 1)
Description: Duration of response(DOR): time from first documentation of objective tumor response (CR/PR) to first documentation of disease progression (PD) or to death due to any cause, whichever occurred first. DOR: calculated for subgroup of participants with confirmed objective tumor response. Intracranial DOR: calculated for participants with confirmed intracranial objective response. CR:disappearance of all non-lymph node target lesions (where all target lesions are recorded with length of 0mm on Target Lesion eCRF). Any pathological lymph node (recorded as target lesion) must have reduction in short axis to <10mm. PR:30% or more decrease in SLD of target lesion, taking as reference baseline SLD. PD:20% or more increase in the SLD of target lesions relative to baseline or smallest SLD (nadir) recorded since first dose. In addition, also demonstrate absolute increase of at least 5mm (>=5mm) relative to baseline or smallest SLD (nadir) recorded since first dose.
Time Frame: From start of study treatment to first documentation of PD or to death due to any cause, whichever occurred first (maximum of 8 years approximately)
Population: DOR analysis set included all ITT participants who had confirmed objective response; intracranial DOR analysis set included all ITT participants who had CNS metastases and achieved confirmed intracranial objective response. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data foe every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Positive Population (Phase 1) | ROS1 Positive Population (Phase 1)
Number analyzed (Participants) | 16 | 6
Participants
  Participants with DOR: number analyzed (Participants) | 10 | 4
  Participants with DOR: <3 Months | 1 | 0
  Participants with DOR: 3 Months to <6 Months | 6 | 0
  Participants with DOR: 6 Months to <9 Months | 0 | 1
  Participants with DOR: 9 Months to <12 Months | 0 | 1
  Participants with DOR: 12 Months to <15 Months | 1 | 0
  Participants with DOR: 15 Months to <18 Months | 0 | 0
  Participants with DOR: 18 Months to <21 Months | 0 | 0
  Participants with DOR: 21 Months to <24 Months | 1 | 0
  Participants with DOR: >=24 Months | 1 | 2
  Participants censored-DOR: number analyzed (Participants) | 6 | 2
  Participants censored-DOR: <3 Months | 0 | 0
  Participants censored-DOR: 3 Months to <6 Months | 0 | 0
  Participants censored-DOR: 6 Months to <9 Months | 0 | 0
  Participants censored-DOR: 9 Months to <12 Months | 0 | 0
  Participants censored-DOR: 12 Months to <15 Months | 0 | 0
  Participants censored-DOR: 15 Months to <18 Months | 0 | 0
  Participants censored-DOR: 18 Months to <21 Months | 0 | 0
  Participants censored-DOR: 21 Months to <24 Months | 0 | 1
  Participants censored-DOR: >=24 Months | 6 | 1
  Participants with intracranial DOR: number analyzed (Participants) | 3 | 0
  Participants with intracranial DOR: <3 Months | 1 | 0
  Participants with intracranial DOR: 3 Months to <6 Months | 0 | 0
  Participants with intracranial DOR: 6 Months to <9 Months | 1 | 0
  Participants with intracranial DOR: 9 Months to <12 Months | 0 | 0
  Participants with intracranial DOR: 12 Months to <15 Months | 1 | 0
  Participants with intracranial DOR: 15 Months to <18 Months | 0 | 0
  Participants with intracranial DOR: 18 Months to <21 Months | 0 | 0
  Participants with intracranial DOR: 21 Months to <24 Months | 0 | 0
  Participants with intracranial DOR: >=24 Months | 0 | 0
  Participants censored- intracranial DOR: number analyzed (Participants) | 11 | 4
  Participants censored- intracranial DOR: <3 Months | 1 | 1
  Participants censored- intracranial DOR: 3 Months to <6 Months | 2 | 0
  Participants censored- intracranial DOR: 6 Months to <9 Months | 0 | 0
  Participants censored- intracranial DOR: 9 Months to <12 Months | 0 | 0
  Participants censored- intracranial DOR: 12 Months to <15 Months | 1 | 0
  Participants censored- intracranial DOR: 15 Months to <18 Months | 0 | 0
  Participants censored- intracranial DOR: 18 Months to <21 Months | 1 | 2
  Participants censored- intracranial DOR: 21 Months to <24 Months | 0 | 0
  Participants censored- intracranial DOR: >=24 Months | 6 | 1

6. Secondary Outcome: Percentage of Participants Achieving Disease Control and Intracranial Disease Control at 12 and 24 Weeks (Phase 1)
Description: Tumor response was evaluated according to RECIST version 1.1, and disease control: confirmed CR, confirmed PR, or stable disease (SD). Intracranial assessment was only performed for participants CNS metastases. CR was defined as disappearance of all non-lymph node target lesions (where all target lesions are recorded with length of 0mm on Target Lesions eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as 30% or more decrease in SLD of target lesions, taking as reference baseline SLD. Progressive disease: 20% or more increase in SLD of target lesions relative to baseline or smallest SLD (nadir) recorded since first dose. In addition to relative increase of 20%, SLD must also demonstrate absolute increase of at least 5mm (>=5mm) relative to baseline or smallest SLD (nadir) recorded since first dose. Results presented here were based on independent central review.
Time Frame: 12 and 24 weeks
Population: The intent-to-treat (ITT) analysis set was used for overall response assessment, and included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922; participants with CNS metastases in the ITT analysis set was used for intracranial response assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ALK Positive Population (Phase 1) | ROS1 Positive Population (Phase 1)
Number analyzed (Participants) | 41 | 12
Percentage of participants
  DCR at Week 12 | 53.7 [37.4 to 69.3] | 58.3 [27.7 to 84.8]
  DCR at Week 24 | 39.0 [24.2 to 55.5] | 50.0 [21.1 to 78.9]
  Intracranial DCR at Week 12: number analyzed (Participants) | 34 | 8
  Intracranial DCR at Week 12 | 50.0 [32.4 to 67.6] | 37.5 [8.5 to 75.5]
  Intracranial DCR at Week 24: number analyzed (Participants) | 34 | 8
  Intracranial DCR at Week 24 | 41.2 [24.6 to 59.3] | 37.5 [8.5 to 75.5]

7. Secondary Outcome: Probability of First Event Being a Central Nervous System (CNS) Progression, Non CNS Progression, or Death (Phase 1)
Description: The probability of the first event being a CNS progression, a non-CNS progression, or death was evaluated with a competing risk approach by estimating cumulative incidence functions (range: 0-1) relative to the analysis set. The time to first event being a Competing Event (either "CNS progression" or "non CNS progression" or "Death") was defined as time from first dose until the date of that specific event. Participants not known to have any of the Competing Events were censored on the date they were last assessed for disease status for PFS. Participants who presented one type of event were counted as a competing cause of failure for the analysis of other type of events. For each type of event, the cumulative incidence function corresponding to the nearest time point preceding 1 year is presented. The results are based on independent central review.
Time Frame: 3 years
Population: The intent-to-treat (ITT) analysis set included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922.
Measure: Number; unit: Probability of events
Groups:
- Phase 1 ITT Population: This reporting group includes all Phase 1 participants in the ITT analysis set.
Arm/Group | Phase 1 ITT Population
Number analyzed (Participants) | 53
Probability of events
  CNS progression | 0.260
  Non CNS progression | 0.352
  Death | 0.060

8. Secondary Outcome: Progression-Free Survival (PFS) (Phase 1)
Description: PFS was defined as the time from the first dose of study treatment to the first documentation of objective PD or to death on study due to any cause, whichever came first. Progressive disease was defined by a 20% or more increase in the SLD of target lesions relative to baseline or the smallest SLD (nadir) recorded since first dose. In addition to the relative increase of 20%, SLD must also demonstrate an absolute increase of at least 5 mm (>= 5 mm) relative to baseline or the smallest SLD (nadir) recorded since the first dose. Results presented here were based on independent central review.
Time Frame: as for outcome 5
Population: PFS analysis set included all participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ALK Positive Population (Phase 1) | ROS1 Positive Population (Phase 1)
Number analyzed (Participants) | 41 | 12
Months | 5.4 [2.7 to 11.8] | 10.1 [1.6 to 33.0]

9. Secondary Outcome: Overall Survival (OS) (Phase 1)
Description: OS was defined as the time from first dose to the date of death due to any cause. For participants still alive at the time of analysis, the OS time was censored on the last date the participants were known to be alive. Estimates of OS and its 95% confidence interval were determined using Kaplan-Meier method.
Time Frame: 3 years
Population: The intent-to-treat (ITT) analysis set included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922. Here, "Number Analyzed" signifies participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ALK Positive Population (Phase 1) | ROS1 Positive Population (Phase 1)
Number analyzed (Participants) | 41 | 12
Months | 22.3 [11.4 to NA] — A large proportion of participants in the analysis set had their OS data censored, and number of participants dead by the cutoff date of this report was small, so it's impossible to derive such summary statistics. | NA [4.7 to NA] — A large proportion of participants in the analysis set had their OS data censored, and number of participants dead by the cutoff date of this report was small, so it's impossible to derive such summary statistics.

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06463922 Following Single Oral Doses (Phase 1)
Description: Maximum observed plasma concentration (Cmax) of PF-06463922 was observed directly from data.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 1 for 25 mg QD and 150 mg QD groups; pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24, 48, 72, 96 and 120 hours post-dose on Day -7 for all other groups.
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 2 | 12 | 16 | 3 | 3 | 3 | 3 | 4
Nanograms per milliliter (ng/mL) | 50.80 (17) | 149.2 (71) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 390 and 423 ng/mL, respectively. | 489.1 (45) | 595.5 (37) | 760.0 (58) | 1201 (19) | 202.2 (57) | 594.9 (27) | 507.2 (51)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06463922 Following Multiple Oral Doses (Phase 1)
Description: Maximum Observed Plasma Concentration (Cmax) of PF-06463922 was observed directly from data.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours post-dose on Cycle 1 Day 15 (24-hour samples not collected for BID groups).
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 16 | 3 | 3 | 3 | 3 | 3
ng/mL | 67.29 (18) | 138.1 (35) | 359.7 (27) | 429.6 (48) | 550.2 (32) | 541.0 (42) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 760 and 1430 ng/mL, respectively. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 370 ng/mL. | 550.0 (23) | 600.5 (27)

12. Secondary Outcome: Time for Cmax (Tmax) of PF-06463922 Following Single Oral Doses (Phase 1)
Description: Tmax of PF-06463922 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 2 | 12 | 16 | 3 | 3 | 3 | 3 | 4
Hours | 1.98 [1.00 to 2.97] | 2.00 [0.50 to 2.05] | 1.25 [0.50 to 2.00] | 1.09 [0.50 to 4.03] | 1.96 [0.517 to 4.33] | 1.05 [1.00 to 3.00] | 2.00 [1.18 to 3.00] | 1.20 [0.50 to 1.97] | 1.23 [1.00 to 2.00] | 2.00 [1.10 to 3.07]

13. Secondary Outcome: Time for Cmax (Tmax) of PF-06463922 Following Multiple Oral Doses (Phase 1)
Description: Tmax of PF-06463922 was observed directly from data as time of first occurrence.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours post-dose on Cycle 1 Day 15 (24-hour samples not collected for BID groups).
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 16 | 3 | 3 | 3 | 3 | 3
Hours | 1.00 [1.00 to 1.08] | 1.00 [1.00 to 2.00] | 2.00 [1.92 to 2.75] | 1.03 [0.50 to 2.00] | 1.13 [1.00 to 4.00] | 1.30 [1.00 to 24.0] | 1.61 [1.22 to 2.00] | 0.50 [0.50 to 0.50] | 0.55 [0.50 to 2.05] | 2.00 [1.00 to 2.00]

14. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time Tau (AUCtau) of PF-06463922 Following Single Oral Doses (Phase 1)
Description: Tau refers to the dosing interval, and it equals to 12 or 24 hours for BID or QD dosing, respectively. AUCtau was determined using linear/log trapezoidal method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 1 for 25 mg QD and 150 mg QD groups; pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, and 24 hours post-dose on Day -7 for all other groups.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 2 | 12 | 16 | 3 | 3 | 3 | 3 | 4
Nanogram*hour/milliliter (ng*hr/mL) | 488.2 (21) | 1387 (35) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 3310 and 3880 ng*hr/mL, respectively. | 3990 (55) | 5110 (28) | 7474 (73) | 11410 (43) | 982.4 (9) | 2996 (20) | 2925 (47)

15. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time Tau (AUCtau) of PF-06463922 Following Multiple Oral Doses (Phase 1)
Description: as for outcome 14
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours post-dose on Cycle 1 Day 15 (24-hour samples not collected for BID groups)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 16 | 3 | 2 | 1 | 3 | 3
ng*hr/mL | 752.1 (26) | 1701 (29) | 3367 (39) | 4107 (53) | 5121 (30) | 6157 (9) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 4480 and 12900 ng*hr/mL, respectively. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 2140 ng*hr/mL. | 3574 (35) | 4058 (33)

16. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06463922 Following Single Oral Doses (Phase 1)
Description: AUCinf was calculated as AUClast + (Clast*/kel), where AUClast was the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel was the rate constant for terminal phase.
Time Frame: as for outcome 10
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 10 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 1 | 2 | 11 | 15 | 3 | 2 | 1 | 4
ng*hr/mL | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 698 ng*hr/mL. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 7210 and 7240 ng*hr/mL, respectively. | 7663 (79) | 8236 (25) | 18340 (61) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 2630 and 3690 ng*hr/mL. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 6860 ng*hr/mL. | 6318 (56)

17. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-06463922 Following Single Oral Doses (Phase 1)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as dose/AUCinf, where AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: as for outcome 10
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | 10 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 1 | 2 | 11 | 15 | 3 | 2 | 1 | 4
Liter/hour (L/hr) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 14.3 L/hr. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 6.91 and 6.94 L/hr, respectively. | 9.788 (79) | 12.14 (25) | 10.90 (61) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 9.48 and 13.3 L/hr, respectively. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 10.9 L/hr. | 15.83 (56)

18. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-06463922 Following Multiple Oral Doses (Phase 1)
Description: as for outcome 17
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours post-dose on Cycle 1 Day 15 (24-hour samples not collected for BID groups)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 16 | 3 | 2 | 1 | 3 | 3
L/hr | 13.27 (26) | 14.72 (29) | 14.84 (39) | 17.66 (48) | 19.52 (30) | 24.37 (9) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 15.5 and 44.6 L/hr, respectively. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 16.3 L/hr. | 20.99 (35) | 22.37 (47)

19. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06463922 Following Single Oral Doses (Phase 1)
Description: Vz/F was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug, and calculated as dose/(AUCinf*kel), where AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time, kel was the rate constant for terminal phase.
Time Frame: as for outcome 10
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | 10 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 1 | 2 | 11 | 15 | 3 | 2 | 1 | 4
Liters (L) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 373 L. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 166 and 307 L, respectively. | 367.9 (54) | 356.3 (39) | 307.8 (41) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 362 and 472 L, respectively. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 410 L. | 378.3 (54)

20. Secondary Outcome: Observed Accumulation Ratio (Rac) of PF-06463922 Following Multiple Oral Doses (Phase 1)
Description: Rac was calculated as Day 15 AUCtau/Day -7 AUCtau or Day 1 AUCtau, where AUCtau was the area under the plasma concentration-time profile from time 0 to time tau (12 and 24 hours for BID and QD dosing regimen, respectively).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours post-dose on Cycle 1 Day 15 (24-hour samples not collected for BID groups)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 3 | 3 | 2 | 12 | 15 | 3 | 2 | 1 | 3 | 3
Ratio | 1.543 (0.075056) | 1.237 (0.20817) | 1.105 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. | 1.121 (0.44575) | 1.071 (0.31138) | 1.000 (0.79137) | 0.6500 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. | NA (NA) — These summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 2.09. | 1.231 (0.35228) | 1.523 (0.29569)

21. Secondary Outcome: Terminal Half-Life of PF-06463922 Following Single Oral Doses (Phase 1)
Description: Terminal plasma half-life was defined as the time measured for the plasma concentration to decrease by one half, and calculated as loge(2)/kel, where kel was the rate constant for terminal phase.
Time Frame: as for outcome 10
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours (hr)
Arm/Group | 10 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 1 | 2 | 11 | 15 | 3 | 2 | 1 | 4
Hours (hr) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 18.0 hr. | 23.70 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. Individual values are 16.6 and 30.8 hr, respectively. | 27.22 (8.2961) | 20.89 (5.0308) | 19.80 (3.3045) | 25.55 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. Individual values are 24.6 and 26.5 hr, respectively. | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 26.0 hr. | 17.18 (5.1874)

22. Secondary Outcome: Steady State Accumulation Ratio (Rss) of PF-06463922 Following Multiple Oral Doses (Phase 1)
Description: Rss was calculated as Day 15 AUCtau/Day -7 AUCinf, where AUCtau was the area under the plasma concentration-time profile from time 0 to time tau (12 and 24 hours for BID and QD dosing regimen, respectively), and AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24 hours post-dose on Cycle 1 Day 15 (24-hour samples not collected for BID groups)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 10 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 1 | 2 | 11 | 14 | 2 | 1 | 1 | 3
Ratio | NA (NA) — These summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 0.993. | 0.5600 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. Individual values are 0.401 and 0.719, respectively. | 0.6131 (0.29021) | 0.6603 (0.18604) | 0.3935 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. Individual values are 0.384 and 0.403, respectively. | NA (NA) — These summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 0.815. | NA (NA) — These summary statistics were not calculated when fewer than 3 participants had reportable values. The individual value is 0.542. | 0.7687 (0.13552)

23. Secondary Outcome: Renal Clearance (CLr) of PF-06463922 (Phase 1)
Description: Renal clearance was calculated as Aetau/AUCtau, where Aetau was the cumulative amount of drug recovered unchanged in urine up to dosing interval tau (24 hours for QD dosing regimen), and AUCtau was the area under the plasma concentration-time profile from time 0 to time tau (24 hours for QD dosing regimen).
Time Frame: 0-4 hours, 4-12 hours and 12-24 hours post-dose on Cycle 1 Day 15
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922. As planned, this parameter was only analyzed for 100 mg QD group. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml/hour
Arm/Group | 100 mg QD (Phase 1)
Number analyzed (Participants) | 3
ml/hour | 61.31 (58)

24. Secondary Outcome: Percent of PF-06463922 Recovered Unchanged in Urine up to Dosing Interval (AEtau%) (Phase 1)
Description: Dosing interval was 24 hours for QD dosing regimen. Aetau% was calculated as 100*Ae24/dose, where Ae24 was the cumulative amount of drug recovered unchanged in urine up to 24 hours post-dose.
Time Frame: 0-4 hours, 4-12 hours and 12-24 hours post-dose on Cycle 1 Day 15
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Percentage of recovered PF-06463922
Arm/Group | 100 mg QD (Phase 1)
Number analyzed (Participants) | 3
Percentage of recovered PF-06463922 | 0.4017 (0.11074)

25. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Midazolam (Phase 1)
Description: Cmax of midazolam was observed directly from data. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflected the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflected the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 9 and 24 hours post-dose on Day -7 and pre-dose, 0.5, 1, 2, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
ng/mL
  Day -7 | 16.06 (42) | 11.56 (48)
  Cycle 1 Day 15 | 9.697 (40) | 5.734 (43)

26. Secondary Outcome: Time for Cmax (Tmax) of Midazolam (Phase 1)
Description: Tmax of midazolam was observed directly from data as time of first occurrence. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflect the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflect the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: as for outcome 25
Population: PK parameter analysis set for midazolam included all participants who received at least 1 dose of midazolam and for which at least 1 midazolam PK parameter of interest was available.
Measure: Median (Full Range); unit: Hours
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
Hours
  Day -7 | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.50]
  Cycle 1 Day 15 | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.533]

27. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Midazolam (Phase 1)
Description: Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) of midazolam was determined using linear/log trapezoidal method. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflect the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflect the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: as for outcome 25
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
ng*hr/mL
  Day -7 | 51.30 (47) | 36.49 (20)
  Cycle 1 Day 15 | 20.43 (18) | 14.44 (25)

28. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Midazolam (Phase 1)
Description: AUCinf was calculated as AUClast + (Clast*/kel), where AUClast was the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel was the rate constant for terminal phase. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflect the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflect the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: as for outcome 25
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
ng*hr/mL
  Day -7: number analyzed (Participants) | 3 | 2
  Day -7 | 54.53 (43) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 42.2 and 46.8 ng*hr/mL, respectively.
  Cycle 1 Day 15 | 21.32 (18) | 16.09 (29)

29. Secondary Outcome: Apparent Oral Clearance (CL/F) of Midazolam (Phase 1)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as dose/AUCinf, where AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflect the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflect the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: as for outcome 25
Population: PK parameter analysis set for midazolam included all participants who received at least 1 dose of midazolam and for which at least 1 midazolam PK parameter of interest was available. Here, 'Number Analyzed' signifies participants evaluable for specified rows
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
L/hr
  Day -7: number analyzed (Participants) | 3 | 2
  Day -7 | 36.68 (43) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 42.7 and 47.4 L/hr, respectively.
  Cycle 1 Day 15 | 93.86 (18) | 124.2 (29)

30. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Midazolam (Phase 1)
Description: Vz/F was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug, and calculated as dose/(AUCinf*kel), where AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time, kel was the rate constant for terminal phase. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflect the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflect the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: as for outcome 25
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
Liters
  Day -7: number analyzed (Participants) | 3 | 2
  Day -7 | 229.0 (7) | NA (NA) — Summary statistics were not calculated when fewer than 3 participants had reportable values. Individual values are 161 and 486 L, respectively.
  Cycle 1 Day 15 | 404.4 (51) | 702.2 (100)

31. Secondary Outcome: Terminal Half-Life of Midazolam (Phase 1)
Description: Terminal plasma half-life was defined as the time measured for the plasma concentration to decrease by one half, and calculated as loge(2)/kel, where kel was the rate constant for terminal phase. Only participants in 25 mg and 150 mg QD groups were given midazolam. Day -7 data reflect the PK assessment before administration of PF-06463922, and Cycle 1 Day 15 data reflect the PK assessment after multiple doses of PF-06463922 were administered.
Time Frame: as for outcome 25
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 25 mg QD (Phase 1) | 150 mg QD (Phase 1)
Number analyzed (Participants) | 3 | 3
Hours
  Day -7: number analyzed (Participants) | 3 | 2
  Day -7 | 4.620 (1.9328) | 5.120 (NA) — Standard deviation was not calculated when fewer than 3 participants had reportable values. Individual values are 2.35 and 7.89 hr, respectively.
  Cycle 1 Day 15 | 3.343 (2.0358) | 5.257 (5.0639)

32. Secondary Outcome: Number of Participants With ALK Mutation Based on Plasma CNA Analysis (Phase 1)
Description: Plasma circulating nucleic acid (CNA) samples were analyzed for ALK kinase domain mutations by digital polymerase chain reaction (PCR) BEAMing technology. Number of participants with one or more ALK mutations is presented.
Time Frame: Screening (up to 28 days)
Population: CNA peripheral blood analysis set included all participants of the ITT analysis set who had at least 1 molecular biomarker assayed.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Positive Population (Phase 1)
Number analyzed (Participants) | 40
Participants | 14

33. Secondary Outcome: Number of Participants With ALK Mutation Based on Tumor Tissue Analysis (Phase 1)
Description: Tumor tissues from archived tissue specimens and/or a de novo biopsy were analyzed for ALK kinase domain mutations. Number of participants with one or more ALK mutations is presented.
Time Frame: Screening (up to 28 days)
Population: Tumor Tissue analysis set included all participants of the ITT analysis set who had at least 1 molecular tumor biomarker assayed from either the screening archival or screening de novo tumor biopsy sample (or both).
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Positive Population (Phase 1)
Number analyzed (Participants) | 40
Participants | 7

34. Secondary Outcome: Number of Participants Who Improved, Worsened or Remained Stable in EORTC QLQ-C30 (Phase 1)
Description: European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ)-C30 (version 3.0) consists of 30 questions assessing 5 functional domains (physical, role, emotional, cognitive and social), global quality of life (QoL), disease/treatment related symptoms (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation and diarrhea), and the perceived financial impact of disease. Each scale was transformed to a range of 0 to 100 using standard EORTC algorithm. For global QoL and functional scales, higher score indicate better performance, and improvement was defined as an increase of at least 10 points, worsening was defined as a decrease of at least 10 points. For symptom scales, higher score indicates worse symptoms, and improvement was defined as a decrease of at least 10 points, worsening was defined as an increase of at least 10 points. All scales which had not improved nor worsened were considered stable.
Time Frame: From start of study treatment until end of treatment (maximum of 8 years approximately)
Population: Patient reported outcome (PRO) evaluable analysis set included all enrolled participants who received at least 1 dose of PF-06463922 and completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 PRO Evaluable Population: This reporting group includes all Phase 1 participants who received at least 1 dose of PF-06463922 and completed a baseline and at least 1 post-baseline PRO assessment.
Arm/Group | Phase 1 PRO Evaluable Population
Number analyzed (Participants) | 43
Participants
  Improved in global QoL | 19
  Stable in global QoL | 13
  Worsened in global QoL | 11
  Improved in physical functioning | 5
  Stable in physical functioning | 29
  Worsened in physical functioning | 9
  Improved in role functioning | 14
  Stable in role functioning | 15
  Worsened in role functioning | 14
  Improved in emotional functioning | 15
  Stable in emotional functioning | 21
  Worsened in emotional functioning | 7
  Improved in cognitive functioning | 8
  Stable in cognitive functioning | 21
  Worsened in cognitive functioning | 14
  Improved in social functioning | 13
  Stable in social functioning | 17
  Worsened in social functioning | 13
  Improved in fatigue | 17
  Stable in fatigue | 19
  Worsened in fatigue | 7
  Improved in nausea and vomiting | 10
  Stable in nausea and vomiting | 32
  worsened in nausea and vomiting | 1
  Improved in pain | 17
  Stable in pain | 16
  Worsened in pain | 10
  Improved in dyspnea | 13
  Stable in dyspnea | 19
  Worsened in dyspnea | 11
  Improved in insomnia | 19
  Stable in insomnia | 17
  Worsened in insomnia | 7
  Improved in appetite loss | 14
  Stable in appetite loss | 27
  Worsened in appetite loss | 2
  Improved in constipation | 10
  Stable in constipation | 28
  Worsened in constipation | 5
  Improved in diarrhea | 9
  Stable in diarrhea | 28
  Worsened in diarrhea | 6
  Improved in financial difficulties | 7
  Stable in financial difficulties | 20
  Worsened in financial difficulties | 16

35. Secondary Outcome: Number of Participants Who Improved, Worsened or Remained Stable in EORTC QLQ-LC13 (Phase 1)
Description: EORTC QLQ-LC13 is the lung cancer module of EORTC QLQ-C30 and includes questions specific to the disease associated symptoms (dyspnea, cough, hemoptysis, and site specific pain), treatment-related symptoms (sore mouth, dysphagia, neuropathy and alopecia), and analgesic use of lung cancer patients. The scale was transformed to a range of 0 to 100 using standard EORTC algorithm. Higher score indicates worse symptoms, and improvement was defined as a decrease of at least 10 points, worsening was defined as an increase of at least 10 points. All scales which had not improved nor worsened were considered stable.
Time Frame: From start of study treatment until end of treatment (maximum of 8 years approximately)
Population: PRO evaluable analysis set included all enrolled participants who received at least 1 dose of PF-06463922 and completed a baseline and at least 1 post-baseline PRO assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 PRO Evaluable Population
Number analyzed (Participants) | 43
Participants
  Improved in dyspnea | 9
  Stable in dyspnea | 23
  Worsened in dyspnea | 11
  Improved in coughing | 23
  Stable in coughing | 12
  Worsened in coughing | 8
  Improved in hemoptysis | 1
  Stable in hemoptysis | 42
  Worsened in hemoptysis | 0
  Improved in sore mouth | 0
  Stable in sore mouth | 40
  Worsened in sore mouth | 3
  Improved in dysphagia | 4
  Stable in dysphagia | 37
  Worsened in dysphagia | 2
  Improved in peripheral neuropathy | 6
  Stable in peripheral neuropathy | 21
  Worsened in peripheral neuropathy | 16
  Improved in alopecia: number analyzed (Participants) | 42
  Improved in alopecia | 4
  Stable in alopecia: number analyzed (Participants) | 42
  Stable in alopecia | 29
  Worsened in alopecia: number analyzed (Participants) | 42
  Worsened in alopecia | 9
  Improved in chest pain | 16
  Stable in chest pain | 22
  Worsened in chest pain | 5
  Improved in arm or shoulder pain | 10
  Stable in arm or shoulder pain | 27
  Worsened in arm or shoulder pain | 6
  Improved in pain in other parts | 20
  Stable in pain in other parts | 12
  Worsened in pain in other parts | 11

36. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Score (Phase 1)
Description: In Phase 1, the MMSE was collected to assess mental status. The MMSE is a 30 item questionnaire that tests 5 areas of cognitive function: orientation, registration, attention and calculation, recall and language. The maximum score is 30 and minimum score is 0. Highest score indicates no cognitive impairment, lowest score indicates severe cognitive impairment. The MMSE was removed under Amendment 6 of the study protocol, and not required for Phase 2, as the tool was not considered meaningful for assessment of cognitive function.
Time Frame: Baseline, Day 1 of Cycle 1-52, and end of treatment (up to 3 years)
Population: MMSE assessment evaluable analysis set included all participants in the safety analysis set (all participants who received at least 1 dose of PF-06463922) who completed a baseline and at least 1 post-baseline assessment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1)
Number analyzed (Participants) | 2 | 3 | 3 | 9 | 16 | 3 | 2 | 2 | 3 | 4
Units on a scale
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 0 | 2 | 7 | 9 | 0 | 0 | 0 | 1 | 1
  Cycle 1 Day 1 | 1.0 (1.41) |  | -0.5 (0.71) | -0.9 (2.27) | 0.8 (1.39) |  |  |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 3 | 1 | 9 | 16 | 3 | 2 | 2 | 2 | 3
  Cycle 2 Day 1 | 2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.3 (0.58) | 2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.3 (1.41) | 0.0 (1.79) | 4.7 (8.08) | 4.0 (4.24) | 0.0 (0.00) | 0.0 (0.00) | -0.3 (1.15)
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 3 | 2 | 8 | 15 | 2 | 2 | 0 | 1 | 3
  Cycle 3 Day 1 | 2.0 (0.00) | 0.3 (0.58) | -0.5 (0.71) | -0.6 (1.85) | 0.2 (1.52) | 5.0 (8.49) | 3.0 (2.83) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.0 (1.00)
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 2 | 2 | 8 | 14 | 3 | 2 | 0 | 1 | 3
  Cycle 4 Day 1 | 5.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.5 (0.71) | 1.5 (2.12) | -1.1 (1.81) | 0.0 (1.47) | 2.0 (6.24) | -0.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.7 (1.15)
  Cycle 5 Day 1: number analyzed (Participants) | 2 | 2 | 2 | 7 | 11 | 3 | 2 | 0 | 1 | 2
  Cycle 5 Day 1 | 0.5 (3.54) | 0.5 (0.71) | 1.5 (2.12) | 0.3 (1.25) | -0.2 (1.72) | 4.7 (8.14) | 0.5 (6.36) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.5 (0.71)
  Cycle 6 Day 1: number analyzed (Participants) | 2 | 2 | 2 | 7 | 11 | 3 | 2 | 0 | 1 | 3
  Cycle 6 Day 1 | 2.5 (2.12) | 0.5 (0.71) | 1.0 (1.41) | -0.4 (2.70) | 0.3 (0.90) | 4.3 (5.86) | 2.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.3 (2.31)
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 2 | 2 | 7 | 12 | 3 | 2 | 0 | 1 | 3
  Cycle 7 Day 1 | 2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.5 (0.71) | 1.5 (2.12) | -0.1 (1.21) | 0.4 (0.90) | 4.7 (8.33) | 3.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.7 (1.15)
  Cycle 8 Day 1: number analyzed (Participants) | 1 | 2 | 2 | 7 | 12 | 3 | 2 | 0 | 1 | 3
  Cycle 8 Day 1 | -4.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.5 (0.71) | 1.5 (2.12) | -0.1 (2.34) | 0.2 (1.34) | 3.0 (7.81) | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 7 | 11 | 2 | 1 | 0 | 0 | 3
  Cycle 9 Day 1 |  | 0.0 (0.00) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.0 (2.31) | 0.3 (2.10) | 6.0 (8.49) | 6.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  | -0.3 (0.58)
  Cycle 10 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 5 | 10 | 2 | 1 | 0 | 1 | 3
  Cycle 10 Day 1 | -5.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.5 (0.71) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00) | -0.1 (0.88) | 6.5 (9.19) | 6.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.7 (1.53)
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 7 | 12 | 2 | 2 | 0 | 1 | 3
  Cycle 11 Day 1 |  | -0.5 (0.71) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.3 (1.70) | -0.2 (1.53) | 7.0 (8.49) | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 12 | 2 | 2 | 0 | 1 | 3
  Cycle 12 Day 1 |  | 0.5 (0.71) |  | -0.6 (2.19) | -0.2 (2.33) | 6.5 (9.19) | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.7 (0.58)
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 10 | 2 | 2 | 0 | 1 | 2
  Cycle 13 Day 1 |  | 0.5 (0.71) |  | 0.8 (1.79) | 0.5 (2.22) | 5.5 (7.78) | 3.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.5 (0.71)
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 6 | 11 | 2 | 2 | 0 | 1 | 3
  Cycle 14 Day 1 |  | 0.5 (0.71) |  | -0.3 (3.20) | 0.3 (0.79) | 6.0 (8.49) | 2.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 15 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 6 | 9 | 0 | 2 | 0 | 1 | 3
  Cycle 15 Day 1 |  | 0.5 (0.71) |  | -1.7 (5.43) | 0.1 (1.36) |  | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.3 (0.58)
  Cycle 16 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 1 | 2 | 0 | 1 | 2
  Cycle 16 Day 1 |  | 0.0 (1.41) |  | -0.2 (2.49) | -0.2 (1.99) | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1.5 (6.36) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 1 | 2 | 0 | 1 | 3
  Cycle 17 Day 1 |  | -2.0 (2.83) |  | 0.6 (1.95) | 0.1 (1.17) | -3.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.3 (1.53)
  Cycle 18 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 1 | 2 | 0 | 0 | 2
  Cycle 18 Day 1 |  | -0.5 (0.71) |  | 0.8 (1.79) | 0.0 (1.73) | -2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.0 (4.24) |  |  | 0.0 (0.00)
  Cycle 19 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 1 | 2 | 0 | 1 | 2
  Cycle 19 Day 1 |  | -0.5 (0.71) |  | 0.8 (1.79) | -0.6 (2.65) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.5 (4.95) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.5 (0.71)
  Cycle 20 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 1 | 2 | 0 | 1 | 2
  Cycle 20 Day 1 |  | 0.0 (0.00) |  | 0.0 (1.41) | 0.7 (2.12) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.5 (0.71)
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 0 | 2 | 0 | 1 | 2
  Cycle 21 Day 1 |  | -0.5 (0.71) |  | 0.0 (1.41) | 0.1 (2.09) |  | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.5 (0.71)
  Cycle 22 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 9 | 1 | 2 | 0 | 1 | 3
  Cycle 22 Day 1 |  | 0.0 (0.00) |  | 0.4 (1.52) | 0.1 (1.45) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.5 (3.54) |  | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.3 (0.58)
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 8 | 1 | 2 | 0 | 1 | 3
  Cycle 23 Day 1 |  | 0.5 (0.71) |  | 0.0 (1.41) | 0.1 (1.81) | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -2.3 (4.04)
  Cycle 24 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 8 | 1 | 2 | 0 | 1 | 2
  Cycle 24 Day 1 |  | 0.5 (0.71) |  | -0.4 (0.89) | 0.6 (0.74) | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 1.5 (4.95) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 25 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 7 | 1 | 2 | 0 | 1 | 2
  Cycle 25 Day 1 |  | 0.0 (0.00) |  | 0.8 (1.79) | -0.9 (2.27) | -2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 2.5 (4.95) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 26 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 8 | 1 | 2 | 0 | 1 | 3
  Cycle 26 Day 1 |  | 0.5 (0.71) |  | 0.8 (1.79) | -0.4 (2.77) | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 2.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.3 (0.58)
  Cycle 27 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 5 | 7 | 1 | 2 | 0 | 1 | 2
  Cycle 27 Day 1 |  | 0.5 (0.71) |  | 0.8 (1.79) | -0.1 (2.67) | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.0 (1.41)
  Cycle 28 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 4 | 7 | 1 | 2 | 0 | 1 | 3
  Cycle 28 Day 1 |  | 0.5 (0.71) |  | 1.0 (2.00) | 0.7 (0.76) | -2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.0 (2.83) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 29 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 4 | 8 | 1 | 2 | 0 | 1 | 3
  Cycle 29 Day 1 |  | -1.5 (2.12) |  | 0.5 (1.73) | 0.1 (1.81) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 30 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 4 | 5 | 1 | 2 | 0 | 1 | 3
  Cycle 30 Day 1 |  | 0.0 (0.00) |  | 0.8 (1.50) | 0.4 (0.55) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.0 (2.83) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -1.0 (1.00)
  Cycle 31 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 3 | 6 | 1 | 2 | 0 | 0 | 3
  Cycle 31 Day 1 |  | 0.5 (0.71) |  | 1.0 (2.65) | 0.7 (0.82) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 3.0 (4.24) |  |  | 0.0 (0.00)
  Cycle 32 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 3 | 5 | 0 | 2 | 0 | 1 | 2
  Cycle 32 Day 1 |  | 0.0 (0.00) |  | 1.3 (2.31) | 0.4 (0.55) |  | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 33 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 3 | 4 | 0 | 2 | 0 | 1 | 2
  Cycle 33 Day 1 |  | 0.0 (0.00) |  | 1.3 (2.31) | 0.5 (0.58) |  | 3.5 (3.54) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 34 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 4 | 0 | 2 | 0 | 1 | 2
  Cycle 34 Day 1 |  | 0.0 (0.00) |  | 0.0 (0.00) | 0.3 (0.50) |  | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00)
  Cycle 35 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 4 | 0 | 2 | 0 | 1 | 1
  Cycle 35 Day 1 |  | 0.5 (0.71) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.3 (0.50) |  | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Cycle 36 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 1
  Cycle 36 Day 1 |  | -0.5 (0.71) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00) |  | 4.0 (4.24) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Cycle 37 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0
  Cycle 37 Day 1 |  | 0.0 (0.00) |  | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00) |  | 3.5 (4.95) |  |  |
  Cycle 38 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0
  Cycle 38 Day 1 |  | 0.0 (0.00) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (0.00) |  | 3.0 (2.83) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |
  Cycle 39 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0
  Cycle 39 Day 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -0.5 (0.71) |  | 3.5 (4.95) |  |  |
  Cycle 40 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
  Cycle 40 Day 1 |  | 0.5 (0.71) |  | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 4.0 (4.24) |  |  |
  Cycle 41 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
  Cycle 41 Day 1 |  | 0.5 (0.71) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 1.5 (6.36) |  |  |
  Cycle 42 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
  Cycle 42 Day 1 |  | -0.5 (0.71) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 4.0 (4.24) |  |  |
  Cycle 43 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Cycle 43 Day 1 |  | 0.0 (0.00) |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  | 4.0 (4.24) |  |  |
  Cycle 44 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
  Cycle 44 Day 1 |  | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  | 3.0 (4.24) |  |  |
  Cycle 45 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 45 Day 1 |  | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  |
  Cycle 46 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 46 Day 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  |  |  |  |
  Cycle 47 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 47 Day 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  |  |  |  |
  Cycle 48 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 48 Day 1 |  | -3.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  |  |  |  |
  Cycle 49 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 49 Day 1 |  | 0.5 (0.71) |  |  |  |  |  |  |  |
  Cycle 50 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 50 Day 1 |  | -3.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  |  |  |  |  |  |
  Cycle 51 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 51 Day 1 |  | -0.5 (0.71) |  |  |  |  |  |  |  |
  Cycle 52 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 52 Day 1 |  | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  |  |  |  |  |  |  |
  End of treatment: number analyzed (Participants) | 1 | 0 | 3 | 1 | 4 | 0 | 0 | 0 | 1 | 1
  End of treatment | -8.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. |  | 0.7 (1.15) | -2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | -2.3 (5.19) |  |  |  | -15.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.

37. Secondary Outcome: Time to Tumor Response (TTR) and Intracranial TTR (Phase 2 and DDI Sub-study)
Description: Time to tumor response (TTR) was defined as the time from the first dose of study treatment to the first documentation of objective tumor response (CR or PR). For participants whose objective response proceeded from PR to CR, the onset of PR was taken as the onset of response. TTR was only calculated for the subgroup of participants with a confirmed objective tumor response. Intracranial TTR was only calculated for participants with confirmed intracranial objective response. CR was defined as the disappearance of all non-lymph node target lesions (where all target lesions are recorded with a length of 0 mm on Target Lesions eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as a 30 % or more decrease in SLD of target lesions, taking as reference the baseline SLD. Results presented here were based on independent central review.
Time Frame: From first dose of study treatment to the first documentation of objective tumor response (CR or PR) (maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: TTR analysis set included all ITT participants who had confirmed objective response; intracranial TTR analysis set included all ITT participants who had CNS metastases and achieved confirmed intracranial objective response. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Median (Full Range); unit: Months
Groups:
- DDI Sub-study: Participants with advanced ALK positive or ROS1-positive NSCLC who were treatment naïve or had any number of prior cancer therapies with or without asymptomatic CNS metastases were administered a single dose of a probe substrate alone on Day -2. Participants were given PF-06463922 100 mg orally QD starting on Cycle1 Day 1 and along with probe substrate on Day 15 Cycle 1.
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 27 | 21 | 34 | 26 | 17 | 18 | 13
Months
  TTR | 1.4 [1.2 to 5.4] | 1.4 [1.2 to 18.0] | 1.4 [1.1 to 16.6] | 2.6 [1.2 to 16.4] | 1.4 [1.2 to 9.3] | 1.4 [1.3 to 29.7] | 1.4 [1.2 to 11.0]
  Intracranial TTR: number analyzed (Participants) | 6 | 10 | 22 | 24 | 16 | 14 | 4
  Intracranial TTR | 2.1 [1.2 to 2.8] | 1.4 [1.2 to 1.5] | 1.4 [1.1 to 5.7] | 1.7 [1.2 to 17.5] | 1.4 [1.2 to 10.6] | 1.4 [1.2 to 28.9] | 2.0 [1.1 to 4.2]

38. Secondary Outcome: Duration of Response (DOR) and Intracranial DOR (Phase 2 and DDI Substudy)
Description: Duration of response(DOR): time from first documentation of objective tumor response (CR/PR) to first documentation of PD or to death due to any cause, whichever occurred first. DOR: calculated for subgroup of participants with confirmed objective tumor response. Intracranial DOR: calculated for participants with confirmed intracranial objective response. CR:disappearance of all non-lymph node target lesions (where all target lesions are recorded with length of 0mm on Target Lesion eCRF). Any pathological lymph node (recorded as target lesion) must have reduction in short axis to <10mm. PR:30% or more decrease in SLD of target lesion, taking as reference baseline SLD. PD:20% or more increase in the SLD of target lesions relative to baseline or smallest SLD (nadir) recorded since first dose. In addition, also demonstrate absolute increase of at least 5mm (>=5mm) relative to baseline or smallest SLD (nadir) recorded since first dose.
Time Frame: From first dose of study treatment to first documentation of PD or to death due to any cause, whichever occurred first (maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: DOR analysis set included all ITT participants who had confirmed objective response; intracranial DOR analysis set included all ITT participants who had CNS metastases and achieved confirmed intracranial objective response. Here, "Number Analyzed" signifies participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 27 | 21 | 34 | 26 | 17 | 18 | 13
Months
  DOR | 17.16 [12.45 to 35.09] | 16.56 [4.20 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 11.10 [5.55 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 15.08 [5.55 to 26.28] | 7.03 [4.17 to 11.01] | 19.61 [11.10 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 5.19 [4.17 to NA] — Upper limit could not be calculated due to insufficient number of participants with events.
  Intra-cranial DOR: number analyzed (Participants) | 6 | 10 | 22 | 24 | 16 | 14 | 4
  Intra-cranial DOR | NA [8.28 to NA] — Median and Upper limit could not be calculated due to insufficient number of participants with events.. | NA [20.99 to NA] — Median and Upper limit could not be calculated due to insufficient number of participants with events. | 37.12 [8.38 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 14.52 [11.07 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 10.32 [6.90 to 14.98] | 17.62 [4.99 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | NA [2.76 to NA] — Median and upper limit could not be calculated due to insufficient number of participants with events.

39. Secondary Outcome: Percentage of Participants Achieving Disease Control and Intracranial Disease Control at Week 12 and 24 (Phase 2 and DDI Substudy)
Description: Tumor response was evaluated according to RECIST version 1.1, and disease control was defined as confirmed CR, confirmed PR, or stable disease (SD). CR was defined as the disappearance of all non-lymph node target lesions (where all target lesions are recorded with a length of 0 mm on Target Lesions eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as a 30 % or more decrease in SLD of target lesions, taking as reference the baseline SLD. SD= when neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD is observed, taking as reference the smallest sum diameters while on study. Intracranial assessment was only performed for participants CNS metastases. Results presented here were based on independent central review.
Time Frame: Weeks 12 and 24
Population: The intent-to-treat (ITT) analysis set was used for overall response assessment, and included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922; participants with CNS metastases in the ITT analysis set was used for intracranial response assessment. Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 30 | 27 | 60 | 65 | 46 | 47 | 32
Percentage of participants
  Disease control rate at Week 12 | 93.3 [77.9 to 99.2] | 85.2 [66.3 to 95.8] | 68.3 [55.0 to 79.7] | 64.6 [51.8 to 76.1] | 50.0 [34.9 to 65.1] | 66.0 [50.7 to 79.1] | 56.3 [37.7 to 73.6]
  Disease control rate at Week 24 | 83.3 [65.3 to 94.4] | 63.0 [42.4 to 80.6] | 51.7 [38.4 to 64.8] | 49.2 [36.6 to 61.9] | 32.6 [19.5 to 48.0] | 48.9 [34.1 to 63.9] | 34.4 [18.6 to 53.2]
  Intra-cranial disease control rate at Week 12: number analyzed (Participants) | 8 | 17 | 33 | 45 | 37 | 25 | 16
  Intra-cranial disease control rate at Week 12 | 87.5 [47.3 to 99.7] | 94.1 [71.3 to 99.9] | 75.8 [57.7 to 88.9] | 75.6 [60.5 to 87.1] | 67.6 [50.2 to 82.0] | 72.0 [50.6 to 87.9] | 56.3 [29.9 to 80.2]
  Intra-cranial disease control rate at Week 24: number analyzed (Participants) | 8 | 17 | 33 | 45 | 37 | 25 | 16
  Intra-cranial disease control rate at Week 24 | 75.0 [34.9 to 96.8] | 70.6 [44.0 to 89.7] | 60.6 [42.1 to 77.1] | 62.2 [46.5 to 76.2] | 48.6 [31.9 to 65.6] | 52.0 [31.3 to 72.2] | 43.8 [19.8 to 70.1]

40. Secondary Outcome: Time to Progression on the Last Prior Therapy (Phase 2)
Description: TTP on the last prior therapy was defined as time from the first dose date of the last prior treatment regimen to the date of progression. Progressive disease was defined by a 20% or more increase in the SLD of target lesions relative to baseline or the smallest SLD (nadir) recorded since first dose. In addition to the relative increase of 20%, SLD must also demonstrate an absolute increase of at least 5 mm (>= 5 mm) relative to baseline or the smallest SLD (nadir) recorded since the first dose.
Time Frame: From first dose of study treatment to the date of progression (maximum of 7.5 years for Phase 2)
Population: ITT analysis set included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922. As planned in SAP, this outcome measure was not analyzed for EXP-1 and EXP-6 groups. Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2)
Number analyzed (Participants) | 27 | 60 | 65 | 46
Months
  Prior systemic therapy before PF-06463922 | 11.5 [7.2 to 19.6] | 12.8 [10.9 to 16.9] | 10.2 [7.6 to 15.9] | 3.7 [2.1 to 6.4]
  Prior ALK+/ROS1+ TKI treatment | 11.5 [7.2 to 19.6] | 13.8 [11.2 to 18.1] | 12.1 [7.9 to 16.4] | 3.7 [2.1 to 6.6]
  Prior systemic therapy other than ALK+/ROS1+ TKI | 19.6 [16.1 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 8.5 [5.0 to 12.6] | 5.0 [3.1 to 10.0] | 5.6 [3.5 to 11.2]

41. Secondary Outcome: Time to Tumor Progression (TTP) and Intracranial TTP (Phase 2 and DDI Substudy)
Description: Time to progression (TTP) was defined as the time from the first dose of study treatment to the first documentation of objective PD. Intracranial TTP was defined as the time from the first dose of study treatment to the date of the first documentation of objective progression of intracranial disease, based on either new brain metastases or progression of existing brain metastases. Progressive disease was defined by a 20% or more increase in the SLD of target lesions relative to baseline or the smallest SLD (nadir) recorded since first dose. In addition to the relative increase of 20%, SLD must also demonstrate an absolute increase of at least 5 mm (>= 5 mm) relative to baseline or the smallest SLD (nadir) recorded since the first dose. Results presented here were based on independent central review.
Time Frame: From first dose of study treatment to the first documentation of objective PD (maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: ITT analysis set was used for TTP determination and included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922; ITT participants with CNS metastases were analyzed for intracranial TTP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 30 | 27 | 60 | 65 | 46 | 47 | 32
Months
  TTP | 17.7 [12.5 to 40.5] | 20.6 [5.5 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 8.2 [5.5 to 12.5] | 8.4 [5.6 to 13.7] | 5.6 [4.0 to 8.3] | 12.5 [8.2 to 26.2] | 5.7 [4.1 to 8.3]
  Intracranial TTP | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | NA [15.0 to NA] — Median and Upper limit could not be calculated due to insufficient number of participants with events. | 22.1 [15.7 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 16.4 [12.7 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | NA [34.5 to NA] — Median and Upper limit could not be calculated due to insufficient number of participants with events. | NA [6.9 to NA] — Median and Upper limit could not be calculated due to insufficient number of participants with events.

42. Secondary Outcome: Probability of First Event Being a Central Nervous System (CNS) Progression, Non CNS Progression, or Death (Phase 2)
Description: Probability of first event being CNS progression, non-CNS progression, or death was evaluated with competing risk approach by estimating cumulative incidence functions (range: 0-1) relative to analysis set. Time to first event being Competing Event (either "CNS progression" or "non CNS progression" or "Death") = time from first dose until date of that specific event. Participants not known to have any of Competing Events were censored on date they were last assessed for disease status for PFS. Participants who presented one type of event were counted as competing cause of failure for analysis of other type of events. For each type of event, cumulative incidence function corresponding to nearest time point preceding 1 year is presented. PD:20% or more increase in SLD of target lesion relative to baseline or smallest SLD (nadir) recorded since first dose. SLD must demonstrate absolute increase of atleast 5mm(>=5 mm) relative to baseline or smallest SLD (nadir) recorded since first dose.
Time Frame: From first dose of study treatment until first event of CNS progression (maximum of 7.5 years for Phase 2)
Population: The ITT analysis set included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922.
Measure: Number; unit: Probability of events
Groups:
- Phase 2 ITT Population: This reporting group includes all Phase 2 participants in the ITT analysis set.
Arm/Group | Phase 2 ITT Population
Number analyzed (Participants) | 274
Probability of events
  CNS progression | 0.179
  Non CNS progression | 0.325
  Death | 0.055

43. Secondary Outcome: Progression-Free Survival (PFS) (Phase 2 and DDI Substudy)
Description: as for outcome 8
Time Frame: From first dose of study treatment to first documentation of objective PD or death due to any cause, whichever came first (maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 30 | 27 | 60 | 65 | 46 | 47 | 32
Months | 16.6 [11.8 to 28.3] | 20.6 [5.5 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 6.9 [5.5 to 11.0] | 7.3 [4.2 to 11.1] | 5.5 [3.9 to 8.2] | 9.9 [5.5 to 21.0] | 5.7 [4.0 to 7.1]

44. Secondary Outcome: Overall Survival (Phase 2 and DDI Substudy)
Description: as for outcome 9
Time Frame: From first dose of study treatment until date of death (maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: ITT analysis set included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 30 | 27 | 60 | 65 | 46 | 47 | 32
Months | NA [NA to NA] — Median and 95% CI could not be calculated due to insufficient number of participants with events. | 52.5 [24.4 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | NA [38.5 to NA] — Median and upper limit could not be calculated due to insufficient number of participants with events. | 18.7 [15.1 to 34.1] | 20.4 [10.5 to 31.6] | 49.7 [21.0 to NA] — Upper limit could not be calculated due to insufficient number of participants with events. | 19.8 [11.1 to NA] — Upper limit could not be calculated due to insufficient number of participants with events.

45. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-06463922 (Phase 2)
Description: Maximum observed plasma concentration (Cmax) of PF-06463922 was observed directly from data.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24, 48, 72, 96 and 120 hours post-dose on Day -7 and pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 15
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922. Here, "Overall Number Analyzed" signifies participants analyzed for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Phase 2 and Japan LIC PK Analysis Set: PK parameters of PF-06463922 were determined for a small subset of Phase 2 participants and Japan LIC. These participants received PF-06463922 100 mg orally QD and were combined into 1 reporting group for PK analysis. Japan LIC was not included in single-dose PK analysis, ie, they did not contribute to Day -7 data.
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 22
ng/mL
  Day -7: number analyzed (Participants) | 19
  Day -7 | 695.2 (40)
  Cycle 1 Day 15 | 576.5 (42)

46. Secondary Outcome: Time for Cmax (Tmax) of PF-06463922 (Phase 2)
Description: Tmax of PF-06463922 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 45
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922. Here, "Number Analyzed" signifies participants analyzed for this outcome measure. Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 22
Hours
  Day -7: number analyzed (Participants) | 19
  Day -7 | 1.15 [0.50 to 4.02]
  Cycle 1 Day 15 | 1.96 [0.50 to 22.7]

47. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06463922 (Phase 2)
Description: as for outcome 16
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24, 48, 72, 96 and 120 hours post-dose on Day -7
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922. Here, 'Overall Number of Participants Analyzed' signifies participants analyzed for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 16
ng*hour/mL | 9088 (35)

48. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time Tau (AUCtau) of PF-06463922 (Phase 2)
Description: Tau refers to the dosing interval, and it equals to 24 hours for QD dosing which was adopted in Phase 2. AUCtau was determined using linear/log trapezoidal method.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Day -7 and pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 15
Population: PK parameter analysis set for PF-06463922 included all enrolled participants who received at least 1 dose of PF-06463922 and had sufficient information to estimate at least one of the PK parameters of interest for PF-06463922. Here, 'Number Analyzed' signifies participants evaluable for specified row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 22
ng*hour/mL
  Day -7: number analyzed (Participants) | 19
  Day -7 | 5308 (36)
  Cycle 1 Day 15 | 5650 (39)

49. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-06463922 (Phase 2)
Description: as for outcome 17
Time Frame: as for outcome 45
Population: as for outcome 48
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 22
Liter/hour
  Day -7: number analyzed (Participants) | 16
  Day -7 | 11.01 (35)
  Cycle 1 Day 15 | 17.70 (39)

50. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06463922 (Phase 2)
Description: as for outcome 19
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24, 48, 72, 96 and 120 hours post-dose on Day -7
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 16
Liters | 351.5 (37)

51. Secondary Outcome: Terminal Half-Life of PF-06463922 (Phase 2)
Description: as for outcome 21
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9, 24, 48, 72, 96 and 120 hours post-dose on Day -7
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 16
Hours | 23.58 (9.3743)

52. Secondary Outcome: Observed Accumulation Ratio (Rac) of PF-06463922 Following Multiple Oral Doses (Phase 2)
Description: Rac was calculated as Day 15 AUCtau/Day -7 AUCtau, where AUCtau was the area under the plasma concentration-time profile from time 0 to time tau (24 hours for QD dosing regimen which was adopted in Phase 2).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 15
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 20
Ratio | 1.082 (0.42701)

53. Secondary Outcome: Steady State Accumulation Ratio (Rss) of PF-06463922 Following Multiple Oral Doses (Phase 2)
Description: Rss was calculated as Day 15 AUCtau/Day -7 AUCinf, where AUCtau was the area under the plasma concentration-time profile from time 0 to time tau (24 hours for QD dosing regimen which was adopted in Phase 2), and AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 9 and 24 hours post-dose on Cycle 1 Day 15
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Phase 2 and Japan LIC PK Analysis Set
Number analyzed (Participants) | 14
Ratio | 0.6577 (0.28627)

54. Secondary Outcome: Number of Participants With ALK Mutation Based on Plasma CNA Analysis (Phase 2)
Description: Plasma CNA samples were analyzed for ALK kinase domain mutations by Next Generation Sequencing (NGS). Number of participants with one or more ALK mutations is presented.
Time Frame: Screening (up to 28 days)
Population: CNA peripheral blood analysis set included all participants of the ITT analysis set who had at least 1 molecular biomarker assayed. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2)
Number analyzed (Participants) | 30 | 26 | 59 | 61 | 46
Participants | 0 | 6 | 8 | 17 | 14

55. Secondary Outcome: Number of Participants With ALK Mutation Based on Tumor Tissue Analysis (Phase 2)
Description: as for outcome 33
Time Frame: Screening (up to 28 days)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2)
Number analyzed (Participants) | 29 | 26 | 58 | 63 | 44
Participants | 0 | 7 | 8 | 12 | 13

56. Secondary Outcome: Number of Participants Who Improved, Worsened or Remained Stable in EORTC QLQ-C30 (Phase 2 and DDI Sub-study)
Description: as for outcome 34
Time Frame: From first dose of study treatment to end of treatment (maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 30 | 26 | 55 | 60 | 43 | 41 | 32
Participants
  Improved in global QoL | 17 | 11 | 18 | 25 | 17 | 19 | 12
  Stable in global QoL | 10 | 12 | 24 | 22 | 16 | 15 | 18
  Worsened in global QoL | 3 | 3 | 13 | 13 | 10 | 6 | 2
  Missing for global QoL | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in physical functioning | 11 | 8 | 13 | 24 | 8 | 11 | 5
  Stable in physical functioning | 13 | 17 | 38 | 24 | 25 | 23 | 23
  Worsened in physical functioning | 6 | 1 | 4 | 12 | 10 | 6 | 4
  Missing for physical functioning | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in role functioning | 12 | 7 | 15 | 25 | 18 | 17 | 10
  Stable in role functioning | 9 | 16 | 33 | 18 | 13 | 17 | 15
  Worsened in role functioning | 9 | 3 | 7 | 17 | 12 | 5 | 7
  Missing for role functioning | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Improved in emotional functioning | 13 | 12 | 13 | 20 | 17 | 16 | 10
  Stable in emotional functioning | 13 | 14 | 32 | 34 | 20 | 22 | 20
  Worsened in emotional functioning | 4 | 0 | 10 | 6 | 6 | 2 | 2
  Missing for emotional functioning | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in cognitive functioning | 9 | 4 | 5 | 12 | 12 | 12 | 9
  Stable in cognitive functioning | 12 | 14 | 36 | 34 | 19 | 20 | 11
  Worsened in cognitive functioning | 9 | 8 | 14 | 14 | 12 | 8 | 12
  Missing for cognitive functioning | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in social functioning | 14 | 7 | 16 | 20 | 11 | 13 | 13
  Stable in social functioning | 11 | 16 | 33 | 29 | 21 | 18 | 13
  Worsened in social functioning | 5 | 3 | 6 | 11 | 11 | 9 | 6
  Missing for social functioning | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in fatigue | 18 | 14 | 22 | 28 | 26 | 16 | 17
  Stable in fatigue | 8 | 11 | 25 | 23 | 9 | 20 | 9
  Worsened in fatigue | 4 | 1 | 8 | 9 | 8 | 4 | 6
  Missing for fatigue | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in nausea and vomiting | 8 | 5 | 10 | 16 | 13 | 10 | 6
  Stable in nausea and vomiting | 22 | 21 | 44 | 39 | 28 | 28 | 24
  Worsened in nausea and vomiting | 0 | 0 | 1 | 5 | 2 | 2 | 2
  Missing for nausea and vomiting | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in pain | 13 | 10 | 20 | 23 | 19 | 21 | 14
  Stable in pain | 10 | 14 | 25 | 28 | 19 | 12 | 13
  Worsened in pain | 7 | 2 | 10 | 9 | 5 | 7 | 5
  Missing for pain | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in dyspnea | 16 | 10 | 10 | 23 | 14 | 14 | 9
  Stable in dyspnea | 10 | 14 | 33 | 22 | 18 | 17 | 15
  Worsened in dyspnea | 4 | 2 | 12 | 15 | 11 | 9 | 8
  Missing for dyspnea | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in insomnia | 20 | 8 | 18 | 30 | 21 | 19 | 12
  Stable in insomnia | 9 | 13 | 28 | 22 | 16 | 18 | 15
  Worsened in insomnia | 1 | 5 | 9 | 8 | 6 | 3 | 5
  Missing for insomnia | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in appetite loss | 14 | 4 | 18 | 29 | 22 | 20 | 10
  Stable in appetite loss | 16 | 22 | 36 | 26 | 21 | 20 | 20
  Worsened in appetite loss | 0 | 0 | 1 | 5 | 0 | 0 | 2
  Missing for appetite loss | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in constipation | 10 | 5 | 9 | 16 | 11 | 13 | 10
  Stable in constipation | 14 | 19 | 33 | 33 | 29 | 22 | 12
  Worsened in constipation | 6 | 2 | 13 | 11 | 3 | 5 | 10
  Missing for constipation | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in diarrhea | 5 | 3 | 10 | 10 | 10 | 8 | 6
  Stable in diarrhea | 18 | 21 | 40 | 39 | 27 | 28 | 21
  Worsened in diarrhea | 7 | 2 | 5 | 11 | 6 | 4 | 5
  Missing for diarrhea | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Improved in financial difficulties | 10 | 6 | 11 | 13 | 10 | 10 | 9
  Stable in financial difficulties | 17 | 19 | 34 | 38 | 22 | 26 | 16
  Worsened in financial difficulties | 3 | 1 | 10 | 9 | 11 | 4 | 7
  Missing for financial difficulties | 0 | 0 | 0 | 0 | 0 | 1 | 0

57. Secondary Outcome: Number of Participants Who Improved, Worsened or Remained Stable in EORTC QLQ-LC13 (Phase 2 and DDI Sub-study)
Description: as for outcome 35
Time Frame: as for outcome 56
Population: Patient reported outcome (PRO) evaluable analysis set included all enrolled participants who received at least 1 dose of PF-06463922 and completed a baseline and at least 1 post-baseline PRO assessment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 30 | 26 | 55 | 60 | 43 | 41 | 32
Participants
  Improved in dyspnea | 11 | 5 | 9 | 21 | 12 | 12 | 6
  Stable in dyspnea | 16 | 18 | 36 | 25 | 21 | 23 | 18
  Worsened in dyspnea | 3 | 3 | 10 | 14 | 9 | 6 | 8
  Missing-dyspnea | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in coughing | 18 | 9 | 22 | 26 | 18 | 17 | 16
  Stable in coughing | 9 | 13 | 26 | 28 | 15 | 18 | 15
  Worsened in coughing | 3 | 4 | 7 | 6 | 9 | 6 | 1
  Missing-coughing | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in hemoptysis | 4 | 0 | 7 | 5 | 5 | 4 | 1
  Stable in hemoptysis | 24 | 25 | 47 | 52 | 34 | 36 | 31
  Worsened in hemoptysis | 2 | 1 | 1 | 3 | 3 | 1 | 0
  Missing-hemoptysis | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in sore mouth | 0 | 2 | 4 | 9 | 2 | 5 | 4
  Stable in sore mouth | 25 | 20 | 44 | 41 | 33 | 28 | 26
  Worsened in sore mouth | 5 | 4 | 7 | 10 | 7 | 8 | 2
  Missing-sore mouth | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in dysphagia | 3 | 1 | 3 | 7 | 4 | 5 | 3
  Stable in dysphagia | 23 | 24 | 46 | 48 | 33 | 30 | 27
  Worsened in dysphagia | 4 | 1 | 6 | 5 | 5 | 6 | 2
  Missing-dysphagia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in peripheral neuropathy | 4 | 5 | 9 | 5 | 6 | 9 | 9
  Stable in peripheral neuropathy | 10 | 13 | 27 | 33 | 22 | 18 | 16
  Worsened in peripheral neuropathy | 16 | 8 | 19 | 22 | 14 | 14 | 7
  Missing-peripheral neuropathy | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in alopecia | 2 | 1 | 2 | 10 | 10 | 9 | 4
  Stable in alopecia | 18 | 22 | 41 | 40 | 24 | 27 | 21
  Worsened in alopecia | 10 | 3 | 12 | 10 | 8 | 5 | 7
  Missing-alopecia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in chest pain | 11 | 7 | 13 | 18 | 14 | 14 | 13
  Stable in chest pain | 17 | 17 | 35 | 33 | 25 | 24 | 17
  Worsened in chest pain | 2 | 2 | 6 | 9 | 3 | 3 | 2
  Missing-chest pain | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Improved in arm or shoulder pain | 10 | 5 | 14 | 14 | 12 | 12 | 9
  Stable in arm or shoulder pain | 15 | 19 | 30 | 36 | 21 | 22 | 19
  Worsened in arm or shoulder pain | 5 | 2 | 11 | 10 | 9 | 7 | 4
  Missing- arm or shoulder pain | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Improved in pain in other parts | 9 | 6 | 17 | 20 | 15 | 17 | 9
  Stable in pain in other parts | 14 | 15 | 23 | 24 | 9 | 18 | 10
  Worsened in pain in other parts | 7 | 5 | 15 | 16 | 17 | 6 | 12
  Missing-Pain in other parts | 0 | 0 | 0 | 0 | 2 | 0 | 1

58. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Phase 1, Phase 2 and DDI Sub-study)
Description: AE: any untoward medical occurrence in clinical investigation participant administered a product or medical device, regardless of causal relationship to study treatment. Treatment-emergent AEs (TEAEs): AEs which occurred for first time during effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs): any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of ability to conduction normal life function). AEs included SAEs and non-serious AEs. Severity was graded as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.Grade1: mild, Grade2: moderate, Grade3: severe, Grade4: Life threatening consequences; urgent intervention indicated, Grade 5: death related to AE.
Time Frame: From first dose of study treatment to end of treatment (maximum of 8 years for Phase 1, maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06463922.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 65 | 46 | 47 | 32
Participants
  AEs (all causality) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 59 | 65 | 46 | 47 | 32
  AEs (treatment-related) | 3 | 3 | 3 | 11 | 16 | 3 | 3 | 1 | 3 | 4 | 30 | 27 | 56 | 61 | 43 | 45 | 31
  SAEs (all causality) | 3 | 2 | 1 | 6 | 10 | 3 | 2 | 2 | 2 | 2 | 15 | 11 | 34 | 31 | 23 | 21 | 13
  SAEs (treatment-related) | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 3 | 0 | 8 | 6 | 6 | 4 | 1
  Grade 3 or 4 (all causality) | 3 | 3 | 0 | 6 | 12 | 3 | 2 | 2 | 1 | 4 | 22 | 22 | 43 | 50 | 36 | 36 | 24
  Grade 3 or 4 (treatment-related) | 2 | 2 | 0 | 3 | 6 | 2 | 0 | 0 | 1 | 3 | 13 | 15 | 31 | 31 | 22 | 25 | 16
  Grade 5 (all causality) | 1 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 1 | 0 | 3 | 3 | 10 | 11 | 9 | 7 | 5
  Grade 5 (treatment-related) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Phase 1, Phase 2 and DDI Sub-study) - Hematology
Description: Hematology evaluation included hemoglobin, platelets, white blood cell, absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils and absolute basophils. Hematology parameters with any abnormalities were reported in this outcome measure.
Time Frame: as for outcome 58
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06463922. Here 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 47 | 32
Participants
  Anemia | 3 | 3 | 3 | 10 | 16 | 3 | 3 | 3 | 3 | 4 | 24 | 22 | 51 | 52 | 35 | 34 | 25
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 1
  Lymphocyte count decreased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 46 | 32
  Lymphocyte count decreased | 2 | 2 | 2 | 7 | 4 | 3 | 3 | 0 | 0 | 2 | 12 | 14 | 30 | 31 | 21 | 26 | 15
  Lymphocyte count increased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 46 | 32
  Lymphocyte count increased | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4 | 3 | 6 | 1 | 1 | 0 | 2
  Neutrophil count decreased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 46 | 32
  Neutrophil count decreased | 1 | 0 | 0 | 4 | 2 | 0 | 1 | 0 | 0 | 1 | 7 | 3 | 8 | 10 | 2 | 7 | 3
  Platelet count decreased | 2 | 2 | 0 | 4 | 5 | 1 | 0 | 0 | 0 | 1 | 8 | 10 | 18 | 12 | 13 | 13 | 8
  White blood cell decreased | 2 | 1 | 0 | 4 | 2 | 2 | 2 | 0 | 0 | 1 | 9 | 5 | 9 | 13 | 8 | 10 | 4

60. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Phase 1, Phase 2 and DDI Sub-study) - Chemistry
Description: Chemistry evaluation included alanine aminotransferase (ALT), alkaline phosphatase, aspartate aminotransferase (AST), blood bilirubin, creatine phosphokinase (CPK), creatinine, gamma-glutamyl transferase (GGT), calcium, sodium, potassium, magnesium, albumin, glucose (non-fasted), albumin, phosphorus or phosphate, serum amylase and lipase.
Time Frame: as for outcome 58
Population: Safety analysis set: all enrolled participants who received at least 1 dose of PF-06463922. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure. 'Number Analyzed': participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 47 | 32
Participants
  ALT increased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 63 | 45 | 47 | 32
  ALT increased | 2 | 1 | 1 | 6 | 9 | 2 | 2 | 0 | 0 | 3 | 13 | 15 | 25 | 25 | 16 | 15 | 10
  Alkaline phosphatase increased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 63 | 45 | 47 | 32
  Alkaline phosphatase increased | 1 | 1 | 3 | 6 | 10 | 3 | 1 | 0 | 2 | 3 | 10 | 13 | 29 | 27 | 25 | 14 | 9
  AST increased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 63 | 45 | 47 | 32
  AST increased | 2 | 2 | 2 | 5 | 8 | 2 | 2 | 0 | 1 | 3 | 16 | 15 | 36 | 33 | 21 | 18 | 11
  Blood bilirubin increased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 63 | 45 | 47 | 32
  Blood bilirubin increased | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 1 | 1
  CPK increased: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 4 | 3 | 0 | 5 | 2
  CPK increased |  |  |  |  | 1 | 1 |  |  | 1 |  | 2 | 1 | 3 | 1 |  | 2 | 1
  Creatinine increased | 3 | 2 | 3 | 10 | 13 | 3 | 3 | 2 | 2 | 3 | 28 | 22 | 40 | 48 | 34 | 37 | 20
  GGT increased: number analyzed (Participants) | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 2 | 2 | 4 | 3 | 1 | 1 | 2 | 1
  GGT increased | 0 |  |  |  | 1 | 0 | 1 |  | 0 | 2 | 1 | 3 | 2 | 1 | 0 | 1 | 0
  Hypercalcemia | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 8 | 4 | 7 | 8 | 4 | 2 | 5
  Hyperglycemia | 3 | 3 | 2 | 7 | 8 | 2 | 1 | 1 | 2 | 1 | 17 | 18 | 37 | 48 | 34 | 31 | 23
  Hyperkalemia | 0 | 1 | 2 | 3 | 6 | 1 | 1 | 1 | 1 | 2 | 11 | 13 | 21 | 13 | 7 | 6 | 5
  Hypermagnesemia: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 59 | 64 | 45 | 47 | 32
  Hypermagnesemia | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 2 | 1 | 4 | 0
  Hypernatremia | 0 | 1 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 1 | 6 | 6 | 9 | 5 | 4 | 5 | 3
  Hypoalbuminemia: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 63 | 45 | 46 | 32
  Hypoalbuminemia | 2 | 1 | 3 | 4 | 7 | 3 | 1 | 1 | 3 | 1 | 19 | 20 | 37 | 43 | 32 | 29 | 18
  Hypocalcemia | 1 | 0 | 1 | 4 | 5 | 2 | 1 | 0 | 0 | 1 | 5 | 5 | 16 | 9 | 6 | 12 | 6
  Hypoglycemia | 0 | 0 | 1 | 3 | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 10 | 9 | 6 | 3 | 6
  Hypokalemia | 0 | 0 | 2 | 4 | 3 | 3 | 1 | 1 | 0 | 2 | 11 | 2 | 10 | 12 | 8 | 14 | 7
  Hypomagnesemia: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 59 | 64 | 45 | 47 | 32
  Hypomagnesemia | 0 | 1 | 2 | 4 | 2 | 3 | 0 | 1 | 1 | 3 | 6 | 9 | 23 | 20 | 16 | 15 | 15
  Hyponatremia | 2 | 1 | 1 | 2 | 4 | 1 | 1 | 0 | 2 | 2 | 7 | 9 | 15 | 23 | 12 | 12 | 10
  Hypophosphatemia: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 59 | 64 | 45 | 47 | 32
  Hypophosphatemia | 1 | 2 | 0 | 3 | 3 | 2 | 1 | 1 | 2 | 1 | 8 | 9 | 23 | 19 | 8 | 15 | 9
  Lipase increased: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 59 | 63 | 45 | 46 | 32
  Lipase increased | 3 | 0 | 0 | 8 | 6 | 0 | 1 | 0 | 2 | 2 | 10 | 7 | 14 | 16 | 15 | 18 | 7
  Serum amylase increased: number analyzed (Participants) | 3 | 3 | 1 | 11 | 16 | 3 | 3 | 3 | 2 | 4 | 30 | 25 | 57 | 63 | 45 | 45 | 32
  Serum amylase increased | 3 | 0 | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 2 | 13 | 6 | 18 | 20 | 11 | 15 | 4

61. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Phase 1, Phase 2 and DDI Sub-study) - Coagulation, Lipids and Urinalysis
Description: Coagulation evaluation included activated partial thromboplastin time, international normalized ratio (INR), and prothrombin time. Lipid evaluation included Cholesterol and triglycerides.
Time Frame: as for outcome 58
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 46 | 32
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 3 | 3 | 3 | 11 | 14 | 3 | 3 | 3 | 3 | 3 | 5 | 5 | 17 | 21 | 15 | 19 | 21
  Activated partial thromboplastin time prolonged | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 3 | 4 | 2
  Cholesterol high: number analyzed (Participants) | 2 | 2 | 2 | 12 | 17 | 2 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 46 | 32
  Cholesterol high | 2 | 2 | 2 | 10 | 16 | 2 | 3 | 3 | 2 | 3 | 30 | 26 | 58 | 64 | 45 | 44 | 31
  Hypertriglyceridemia: number analyzed (Participants) | 1 | 2 | 2 | 12 | 17 | 2 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 64 | 45 | 46 | 32
  Hypertriglyceridemia | 0 | 2 | 2 | 11 | 16 | 2 | 3 | 2 | 1 | 3 | 30 | 26 | 56 | 61 | 45 | 43 | 31
  INR increased: number analyzed (Participants) | 3 | 3 | 3 | 11 | 14 | 3 | 3 | 3 | 3 | 3 | 6 | 10 | 20 | 31 | 20 | 26 | 24
  INR increased | 2 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 6 | 2 | 7 | 3
  Prothrombin time: number analyzed (Participants) | 3 | 3 | 3 | 11 | 14 | 3 | 3 | 3 | 3 | 3 | 6 | 8 | 18 | 29 | 21 | 21 | 21
  Prothrombin time | 2 | 1 | 1 | 3 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 6 | 6 | 3 | 6 | 6

62. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-defined Criteria (Phase 1, Phase 2 and DDI Sub-study)
Description: Blood pressure (BP), including systolic BP (SBP) and diastolic BP (DBP), and pulse rate were recorded in sitting position. Body weight was also measured.
Time Frame: as for outcome 58
Population: Safety analysis set: all enrolled participants who received at least 1 dose of PF-06463922. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure. 'Number Analyzed': participants evaluable for specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 65 | 45 | 46 | 32
Participants
  Increase in sitting SBP >=40 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Increase in sitting SBP >=40 mmHg | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 9 | 7 | 10 | 10 | 5 | 4 | 4
  Increase in sitting SBP >=60 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Increase in sitting SBP >=60 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Decrease in sitting SBP >=40 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Decrease in sitting SBP >=40 mmHg | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 2 | 2 | 3 | 1
  Decrease in sitting SBP >=60 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Decrease in sitting SBP >=60 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Increase in sitting DBP >=20 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Increase in sitting DBP >=20 mmHg | 0 | 2 | 0 | 0 | 7 | 3 | 1 | 0 | 1 | 0 | 11 | 12 | 21 | 15 | 15 | 12 | 7
  Increase in sitting DBP >=40 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Increase in sitting DBP >=40 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 0
  Decrease in sitting DBP >=20 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Decrease in sitting DBP >=20 mmHg | 2 | 1 | 0 | 5 | 3 | 2 | 2 | 0 | 1 | 2 | 9 | 5 | 15 | 10 | 10 | 9 | 8
  Decrease in sitting DBP >=40 mmHg: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 45 | 44 | 32
  Decrease in sitting DBP >=40 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Sitting pulse rate <50 bpm | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 1 | 0 | 2 | 2
  Sitting pulse rate >120 bpm | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 9 | 4 | 2 | 3
  Increase in sitting pulse rate >=30 bpm: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 44 | 44 | 32
  Increase in sitting pulse rate >=30 bpm | 0 | 1 | 0 | 2 | 7 | 1 | 0 | 0 | 0 | 1 | 0 | 7 | 14 | 19 | 17 | 17 | 8
  Decrease in sitting pulse rate >=30 bpm: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 60 | 65 | 44 | 44 | 32
  Decrease in sitting pulse rate >=30 bpm | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 11 | 2 | 8 | 7 | 3 | 5 | 4
  Increase in weight: 10% to <20%: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 58 | 61 | 44 | 43 | 32
  Increase in weight: 10% to <20% | 1 | 0 | 0 | 8 | 6 | 2 | 2 | 0 | 0 | 0 | 9 | 14 | 17 | 15 | 11 | 14 | 9
  Increase in weight: >=20%: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 58 | 61 | 44 | 43 | 32
  Increase in weight: >=20% | 0 | 2 | 1 | 1 | 5 | 1 | 0 | 0 | 1 | 1 | 12 | 2 | 10 | 16 | 9 | 9 | 3
  Decrease in weight >=10%: number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 26 | 58 | 61 | 44 | 43 | 32
  Decrease in weight >=10% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 3 | 4 | 2 | 2 | 1

63. Secondary Outcome: Number of Participants With Maximum Decrease From Baseline Greater Than or Equal to 20 Percent in Left Ventricular Ejection Fraction (LVEF) (Phase 1, Phase 2 and DDI Sub-study)
Description: Left Ventricular Ejection Fraction (LVEF) was determined by echocardiogram. Baseline was defined as the measurement prior to the first dose of study treatment.
Time Frame: as for outcome 58
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06463922.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 65 | 46 | 47 | 32
Participants | 1 | 0 | 1 | 3 | 5 | 2 | 1 | 0 | 0 | 2 | 4 | 2 | 13 | 14 | 3 | 5 | 2

64. Secondary Outcome: Number of Participants With Absolute Values and Change From Baseline in QTcF Meeting Pre-defined Criteria (Phase 1, Phase 2 and DDI Sub-study)
Description: Triplicate 12-lead electrocardiograms (ECGs) were performed approximately 2 minutes apart to determine mean QTc interval (QT interval corrected for heart rate). QT interval was corrected for heart rate using Fridericia's formula to provide QTcF. Absolute values and changes from baseline were summarized according to pre-defined criteria. Baseline was defined as the last evaluation on or prior to the first dose of study treatment.
Time Frame: as for outcome 58
Population: The safety analysis set included all enrolled participants who received at least 1 dose of PF-06463922.
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Sub-study
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 17 | 3 | 3 | 3 | 3 | 4 | 30 | 27 | 60 | 65 | 46 | 47 | 32
Participants
  QTcF: 450 to <480 msec | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 5 | 8 | 11 | 9 | 13 | 9 | 7
  QTcF: 480 to <500 msec | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 1 | 1
  QTcF: >=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
  QTcF Increase: 30 to <60 msec | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 1 | 0 | 1 | 10 | 8 | 18 | 20 | 7 | 12 | 7
  QTcF: >=60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 1

65. Secondary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior (Phase 2)
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) was used to analyze participants' suicidal ideation and behavior, and it is a unique, simple and short method of assessing both behavior and ideation that tracks all suicidal events and provides a summary of suicidality. It assesses the lethality of attempts and other features of ideation (frequency, duration, controllability, reasons for ideation and deterrents), all of which are significantly predictive of completed suicide. Maximum score of 4 or 5 indicates maximum suicidal ideation and minimum score of "0" indicates no suicidal ideation.
Time Frame: From first dose of study treatment to end of treatment (maximum of 7.5 years for Phase 2)
Population: PRO evaluable analysis set included all enrolled participants who received study treatment, had a baseline test assessment and at least 1 on-study test assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 26 | 24 | 52 | 43 | 30 | 25
Participants
  Suicidal ideation | 1 | 0 | 2 | 1 | 1 | 2
  Suicidal behavior | 0 | 0 | 0 | 0 | 0 | 1

66. Secondary Outcome: Change From Baseline in Total Scores for Beck Depression Inventory (BDI)-II (Mood Assessment) (Phase 2)
Description: The Beck Depression Inventory (BDI)-II is a 21-item self-report scale, with each item rated by participants on a 4-point scale (ranging from 0-3, where 0 indicated lowest depression and 3 indicated severe depression). The scale includes items capturing mood, (loss of pleasure, sadness, and irritability), suicidal ideation, and cognitive signs (punitive thoughts, self-criticism, self-dislike, pessimism, and poor concentration) as well as somatic signs (appetite, sleep, fatigue and libido). Scores were obtained by adding up the total points from the series of answers. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs are as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Time Frame: Baseline, Day 1 of Cycles 2-5, Day 1 of every other cycle from Cycle 6, and end of treatment (up to 3 years)
Population: PRO evaluable analysis set included all enrolled participants who received study treatment, had a baseline test assessment and at least 1 on-study test assessment. Here, 'Number Analyzed' signifies participants evaluable for specified row.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 24 | 24 | 53 | 41 | 28 | 26
Units on a scale
  Cycle 2 Day 1 | -2.59 [-4.82 to -0.37] | -3.27 [-5.52 to -1.01] | -2.26 [-3.77 to -0.76] | -2.17 [-3.89 to -0.46] | -1.52 [-3.60 to 0.56] | -2.43 [-4.57 to -0.29]
  Cycle 3 Day 1 | -3.34 [-5.57 to -1.12] | -3.18 [-5.43 to -0.93] | -3.03 [-4.55 to -1.51] | -3.10 [-4.85 to -1.35] | -0.46 [-2.61 to 1.69] | -1.24 [-3.37 to 0.90]
  Cycle 4 Day 1 | -3.84 [-6.07 to -1.62] | -4.10 [-6.38 to -1.82] | -2.59 [-4.14 to -1.05] | -1.95 [-3.72 to -0.19] | -1.19 [-3.38 to 1.01] | -1.94 [-4.12 to 0.24]
  Cycle 5 Day 1 | -4.47 [-6.69 to -2.24] | -3.96 [-6.27 to -1.66] | -2.75 [-4.33 to -1.16] | -3.03 [-4.82 to -1.25] | -1.51 [-3.74 to 0.72] | -1.25 [-3.46 to 0.95]
  Cycle 6 Day 1 | -3.51 [-5.73 to -1.28] | -4.25 [-6.56 to -1.94] | -3.31 [-4.90 to -1.72] | -3.79 [-5.61 to -1.98] | -0.42 [-2.64 to 1.81] | -0.29 [-2.54 to 1.96]
  Cycle 8 Day 1 | -4.17 [-6.41 to -1.92] | -4.86 [-7.23 to -2.50] | -2.26 [-3.86 to -0.66] | -4.06 [-5.90 to -2.22] | -1.09 [-3.34 to 1.17] | 0.17 [-2.10 to 2.45]
  Cycle 10 Day 1 | -3.09 [-5.38 to -0.80] | -4.92 [-7.28 to -2.55] | -1.94 [-3.54 to -0.34] | -4.27 [-6.14 to -2.39] | -2.97 [-5.29 to -0.66] | -0.19 [-2.60 to 2.22]
  Cycle 12 Day 1 | -3.95 [-6.30 to -1.61] | -5.60 [-7.97 to -3.24] | -0.72 [-2.40 to 0.95] | -4.80 [-6.83 to -2.77] | -1.94 [-4.29 to 0.42] | -1.40 [-3.81 to 1.01]
  Cycle 14 Day 1 | -3.81 [-6.18 to -1.43] | -5.80 [-8.35 to -3.25] | -2.58 [-4.41 to -0.76] | -4.29 [-6.41 to -2.17] | -1.73 [-4.40 to 0.94] | -0.08 [-2.59 to 2.42]
  Cycle 16 Day 1 | -1.75 [-4.40 to 0.89] | -4.61 [-7.51 to -1.71] | -2.15 [-4.35 to 0.06] | -4.65 [-6.90 to -2.41] | -2.22 [-5.50 to 1.07] | 0.03 [-2.65 to 2.71]
  Cycle 18 Day 1 | -4.49 [-7.49 to -1.49] | -7.02 [-10.59 to -3.46] | -1.96 [-4.22 to 0.31] | -2.86 [-5.21 to -0.51] | -1.11 [-8.25 to 6.03] | 1.88 [-1.66 to 5.41]
  Cycle 20 Day 1: number analyzed (Participants) | 24 | 24 | 53 | 41 | 0 | 26
  Cycle 20 Day 1 | -5.01 [-8.55 to -1.46] | -5.17 [-9.06 to -1.29] | -1.82 [-4.70 to 1.06] | -3.63 [-6.31 to -0.95] |  | 1.88 [-1.66 to 5.41]
  Cycle 22 Day 1: number analyzed (Participants) | 24 | 24 | 53 | 41 | 0 | 26
  Cycle 22 Day 1 | -2.93 [-6.79 to 0.94] | -4.63 [-9.00 to -0.26] | -2.36 [-5.68 to 0.96] | -5.50 [-8.87 to -2.12] |  | -2.39 [-6.73 to 1.94]
  Cycle 24 Day 1: number analyzed (Participants) | 24 | 24 | 53 | 41 | 0 | 26
  Cycle 24 Day 1 | -7.31 [-11.66 to -2.96] | -5.63 [-10.00 to -1.26] | -2.88 [-7.04 to 1.28] | -3.89 [-8.10 to 0.32] |  | 2.27 [-2.06 to 6.61]
  Cycle 26 Day 1: number analyzed (Participants) | 24 | 0 | 53 | 41 | 0 | 0
  Cycle 26 Day 1 | -5.50 [-10.67 to -0.33] |  | -3.03 [-10.01 to 3.95] | -4.30 [-11.31 to 2.70] |  |
  End of treatment | -4.77 [-9.23 to -0.32] | -0.73 [-5.61 to 4.15] | -2.55 [-5.28 to 0.18] | -3.22 [-5.49 to -0.95] | 0.74 [-2.70 to 4.17] | -2.08 [-5.65 to 1.50]

67. Secondary Outcome: Change From Baseline in Total Scores for Detection Test (Cognitive Function Assessment) (Phase 2)
Description: The Detection Test is a measure of psychomotor function and uses a well validated simple reaction time paradigm with playing card stimuli. In this test, the on-screen instructions ask: "Has the card turned over?". A playing card is presented face down in the center of the screen. The card flips over so it is face up. As soon as the card flips over the participant must press "Yes". The participant is encouraged to work as quickly as they can and be as accurate as possible. The speed and accuracy of each response are recorded and mean of the log10 transformed reaction times for correct responses is calculated. Lower values of least square mean change from baseline indicate performance decline. Upper limit of 95% confidence interval of -0.00 or lower indicate statistically significant decline of performance over baseline at that cycle.
Time Frame: Baseline, Day 1 of Cycles 2-5, Day 1 of every other cycle from Cycle 6, and end of treatment (up to 3 years)
Population: as for outcome 66
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 24 | 26 | 50 | 46 | 38 | 29
Units on a scale
  Cycle 2 Day 1 | 0.01 [-0.04 to 0.05] | 0.04 [-0.01 to 0.08] | -0.01 [-0.04 to 0.02] | 0.02 [-0.01 to 0.05] | -0.02 [-0.05 to 0.02] | 0.01 [-0.03 to 0.05]
  Cycle 3 Day 1 | -0.01 [-0.05 to 0.03] | 0.01 [-0.03 to 0.05] | 0.01 [-0.02 to 0.04] | -0.01 [-0.04 to 0.02] | -0.01 [-0.05 to 0.02] | -0.01 [-0.05 to 0.03]
  Cycle 4 Day 1 | 0.03 [-0.02 to 0.07] | 0.00 [-0.04 to 0.04] | -0.03 [-0.06 to 0.00] | -0.02 [-0.05 to 0.01] | -0.04 [-0.07 to -0.00] | -0.01 [-0.06 to 0.03]
  Cycle 5 Day 1 | -0.01 [-0.05 to 0.03] | -0.01 [-0.06 to 0.03] | -0.00 [-0.03 to 0.03] | 0.00 [-0.03 to 0.03] | -0.04 [-0.08 to -0.01] | -0.04 [-0.08 to 0.00]
  Cycle 6 Day 1 | -0.03 [-0.07 to 0.01] | 0.01 [-0.03 to 0.06] | -0.02 [-0.05 to 0.01] | -0.00 [-0.04 to 0.03] | -0.01 [-0.05 to 0.02] | -0.02 [-0.07 to 0.02]
  Cycle 8 Day 1 | -0.02 [-0.06 to 0.02] | 0.00 [-0.04 to 0.05] | -0.02 [-0.05 to 0.01] | -0.03 [-0.06 to 0.01] | -0.04 [-0.07 to 0.00] | 0.00 [-0.04 to 0.05]
  Cycle 10 Day 1 | -0.02 [-0.06 to 0.02] | 0.03 [-0.01 to 0.08] | -0.02 [-0.06 to 0.01] | -0.01 [-0.05 to 0.02] | -0.05 [-0.09 to -0.01] | -0.04 [-0.08 to 0.01]
  Cycle 12 Day 1 | -0.04 [-0.08 to 0.01] | -0.00 [-0.05 to 0.04] | -0.02 [-0.06 to 0.02] | -0.03 [-0.06 to 0.01] | -0.08 [-0.13 to -0.04] | -0.01 [-0.05 to 0.04]
  Cycle 14 Day 1 | 0.02 [-0.04 to 0.07] | 0.02 [-0.03 to 0.08] | -0.05 [-0.09 to -0.01] | -0.04 [-0.08 to -0.00] | -0.02 [-0.07 to 0.04] | 0.01 [-0.05 to 0.06]
  Cycle 16 Day 1 | -0.03 [-0.09 to 0.03] | 0.01 [-0.05 to 0.07] | 0.02 [-0.03 to 0.07] | -0.03 [-0.08 to 0.01] | -0.04 [-0.14 to 0.06] | -0.01 [-0.07 to 0.06]
  Cycle 18 Day 1 | 0.09 [0.01 to 0.18] | -0.02 [-0.09 to 0.05] | -0.03 [-0.09 to 0.02] | -0.06 [-0.11 to -0.01] | -0.09 [-0.23 to 0.04] | -0.01 [-0.08 to 0.05]
  Cycle 20 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 20 Day 1 | 0.07 [-0.03 to 0.17] | 0.02 [-0.06 to 0.09] | 0.01 [-0.06 to 0.08] | -0.09 [-0.16 to -0.03] |  | -0.03 [-0.11 to 0.04]
  Cycle 22 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 22 Day 1 | -0.02 [-0.12 to 0.08] | -0.02 [-0.10 to 0.07] | 0.00 [-0.08 to 0.08] | -0.08 [-0.16 to 0.00] |  | -0.05 [-0.13 to 0.03]
  Cycle 24 Day 1: number analyzed (Participants) | 24 | 0 | 0 | 46 | 0 | 0
  Cycle 24 Day 1 | 0.03 [-0.11 to 0.16] |  |  | -0.06 [-0.20 to 0.07] |  |
  End of treatment | -0.04 [-0.13 to 0.04] | -0.01 [-0.10 to 0.08] | -0.02 [-0.08 to 0.04] | -0.05 [-0.10 to -0.00] | -0.07 [-0.14 to -0.01] | -0.05 [-0.12 to 0.03]

68. Secondary Outcome: Change From Baseline in Total Scores for Identification Test (Cognitive Function Assessment) (Phase 2)
Description: The Identification Test is a measure of visual attention and uses a well validated choice reaction time paradigm with playing card stimuli. In this task, the playing cards are all red or black jokers. The on-screen instructions ask: "Is the card red?". A playing card is presented face down in the center of the screen. The card flips over so it is face up. As soon as it flips over the participant must decide whether the card is red or not. If it is red the participant should press "Yes", and if it is not red the participant should press "No". The participant is encouraged to work as quickly and accurately as possible. The speed and accuracy of each response are recorded and mean of the log10 transformed reaction times for correct responses is calculated. Lower values of least square mean change from baseline indicate performance decline. Upper limit of 95% confidence interval of -0.00 or lower indicate statistically significant decline of performance over baseline at that cycle.
Time Frame: Baseline, Day 1 of Cycles 2-5, Day 1 of every other cycle from Cycle 6, and end of treatment (up to 3 years)
Population: as for outcome 66
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 24 | 26 | 50 | 46 | 38 | 29
Units on a scale
  Cycle 2 Day 1 | -0.02 [-0.05 to 0.01] | -0.02 [-0.05 to 0.01] | -0.01 [-0.03 to 0.00] | -0.01 [-0.03 to 0.01] | -0.02 [-0.04 to 0.01] | -0.01 [-0.04 to 0.02]
  Cycle 3 Day 1 | -0.01 [-0.04 to 0.02] | -0.01 [-0.04 to 0.02] | -0.02 [-0.04 to 0.00] | -0.02 [-0.04 to 0.00] | -0.02 [-0.05 to 0.00] | -0.01 [-0.04 to 0.02]
  Cycle 4 Day 1 | -0.02 [-0.05 to 0.01] | -0.01 [-0.04 to 0.01] | -0.02 [-0.04 to 0.00] | -0.03 [-0.05 to -0.01] | -0.05 [-0.08 to -0.03] | -0.02 [-0.04 to 0.01]
  Cycle 5 Day 1 | -0.03 [-0.06 to -0.00] | -0.02 [-0.05 to 0.01] | -0.03 [-0.05 to -0.00] | -0.02 [-0.04 to 0.01] | -0.05 [-0.07 to -0.02] | -0.02 [-0.05 to 0.00]
  Cycle 6 Day 1 | -0.04 [-0.07 to -0.01] | -0.02 [-0.05 to 0.01] | -0.02 [-0.04 to 0.00] | -0.03 [-0.06 to -0.01] | -0.03 [-0.06 to -0.01] | -0.03 [-0.06 to -0.00]
  Cycle 8 Day 1 | -0.03 [-0.06 to -0.00] | -0.02 [-0.05 to 0.01] | -0.03 [-0.05 to -0.01] | -0.03 [-0.05 to -0.01] | -0.05 [-0.07 to -0.02] | -0.03 [-0.06 to 0.00]
  Cycle 10 Day 1 | -0.03 [-0.06 to 0.00] | -0.01 [-0.04 to 0.02] | -0.03 [-0.05 to -0.01] | -0.02 [-0.05 to 0.00] | -0.05 [-0.08 to -0.02] | -0.03 [-0.06 to 0.00]
  Cycle 12 Day 1 | -0.05 [-0.08 to -0.02] | -0.04 [-0.07 to -0.01] | -0.04 [-0.06 to -0.01] | -0.04 [-0.07 to -0.01] | -0.06 [-0.09 to -0.03] | -0.03 [-0.06 to 0.00]
  Cycle 14 Day 1 | -0.04 [-0.08 to 0.00] | -0.04 [-0.07 to -0.00] | -0.03 [-0.06 to -0.00] | -0.04 [-0.07 to -0.01] | -0.04 [-0.08 to -0.00] | -0.02 [-0.06 to 0.02]
  Cycle 16 Day 1 | -0.09 [-0.13 to -0.05] | -0.00 [-0.04 to 0.04] | -0.03 [-0.07 to 0.01] | -0.03 [-0.06 to 0.01] | -0.07 [-0.13 to 0.00] | -0.06 [-0.10 to -0.01]
  Cycle 18 Day 1 | -0.01 [-0.06 to 0.05] | -0.05 [-0.09 to 0.00] | -0.04 [-0.08 to 0.00] | -0.07 [-0.10 to -0.03] | -0.19 [-0.29 to -0.09] | -0.01 [-0.05 to 0.04]
  Cycle 20 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 20 Day 1 | -0.03 [-0.10 to 0.04] | -0.01 [-0.06 to 0.04] | -0.03 [-0.08 to 0.02] | -0.10 [-0.15 to -0.06] |  | -0.03 [-0.08 to 0.02]
  Cycle 22 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 22 Day 1 | 0.04 [-0.03 to 0.11] | -0.01 [-0.07 to 0.05] | -0.06 [-0.11 to 0.00] | -0.05 [-0.11 to 0.00] |  | -0.08 [-0.14 to -0.03]
  Cycle 24 Day 1: number analyzed (Participants) | 24 | 0 | 0 | 46 | 0 | 0
  Cycle 24 Day 1 | 0.08 [-0.01 to 0.18] |  |  | -0.06 [-0.15 to 0.04] |  |
  End of treatment | -0.07 [-0.13 to -0.02] | -0.03 [-0.10 to 0.03] | -0.02 [-0.06 to 0.02] | -0.03 [-0.06 to 0.01] | -0.09 [-0.14 to -0.05] | -0.06 [-0.11 to -0.01]

69. Secondary Outcome: Change From Baseline in Total Scores for One Back Test (Cognitive Function Assessment) (Phase 2)
Description: The One Back Test is a measure of working memory and uses a well validated n back paradigm with playing cards. In this task, the on-screen instructions ask: "Is the previous card the same?". A playing card is presented in the center of the screen. The participant must decide whether the card is the same as the previous card. If it is the same the participant should press "Yes", and if not press "No". The participant is encouraged to work as quickly and accurately as possible. The speed and accuracy of each response are recorded, mean of the log10 transformed reaction times for correct responses is used to demonstrate speed of performance, and the arcsine transformation of the square root of the proportion of correct responses is used to demonstrate accuracy. Lower values of least square mean change from baseline indicate performance decline. Upper limit of 95% confidence interval of -0.00 or lower indicate statistically significant decline of performance over baseline at that cycle.
Time Frame: Baseline, Day 1 of Cycles 2-5, Day 1 of every other cycle from Cycle 6, and end of treatment (up to 3 years)
Population: as for outcome 66
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 24 | 26 | 50 | 46 | 38 | 29
Units on a scale
  Cycle 2 Day 1 | 0.01 [-0.02 to 0.05] | 0.02 [-0.01 to 0.05] | 0.02 [0.00 to 0.05] | 0.01 [-0.01 to 0.04] | 0.02 [-0.01 to 0.05] | 0.01 [-0.02 to 0.04]
  Cycle 3 Day 1 | 0.06 [0.02 to 0.09] | 0.01 [-0.02 to 0.05] | 0.01 [-0.01 to 0.04] | 0.01 [-0.02 to 0.03] | -0.01 [-0.04 to 0.02] | -0.00 [-0.04 to 0.03]
  Cycle 4 Day 1 | 0.04 [0.01 to 0.08] | 0.03 [-0.00 to 0.06] | 0.02 [-0.01 to 0.04] | -0.01 [-0.04 to 0.01] | -0.02 [-0.05 to 0.01] | -0.01 [-0.05 to 0.02]
  Cycle 5 Day 1 | 0.02 [-0.01 to 0.06] | 0.03 [-0.00 to 0.07] | 0.03 [0.00 to 0.05] | -0.01 [-0.04 to 0.02] | -0.02 [-0.05 to 0.01] | 0.02 [-0.01 to 0.05]
  Cycle 6 Day 1 | 0.03 [-0.01 to 0.06] | 0.03 [-0.00 to 0.07] | 0.03 [0.01 to 0.06] | 0.01 [-0.02 to 0.04] | -0.00 [-0.03 to 0.03] | 0.01 [-0.03 to 0.04]
  Cycle 8 Day 1 | 0.03 [-0.01 to 0.06] | 0.02 [-0.02 to 0.06] | 0.03 [0.00 to 0.05] | 0.01 [-0.02 to 0.03] | -0.01 [-0.04 to 0.02] | 0.01 [-0.02 to 0.05]
  Cycle 10 Day 1 | 0.07 [0.03 to 0.11] | 0.03 [-0.00 to 0.07] | 0.03 [0.00 to 0.05] | 0.02 [-0.01 to 0.05] | -0.01 [-0.05 to 0.02] | 0.01 [-0.02 to 0.05]
  Cycle 12 Day 1 | 0.05 [0.01 to 0.08] | 0.01 [-0.03 to 0.05] | 0.02 [-0.01 to 0.05] | 0.01 [-0.02 to 0.04] | -0.00 [-0.04 to 0.03] | 0.03 [-0.01 to 0.07]
  Cycle 14 Day 1 | 0.00 [-0.05 to 0.05] | 0.03 [-0.01 to 0.07] | 0.03 [-0.01 to 0.07] | -0.00 [-0.04 to 0.03] | 0.01 [-0.04 to 0.06] | 0.02 [-0.03 to 0.07]
  Cycle 16 Day 1 | 0.03 [-0.03 to 0.08] | 0.05 [-0.01 to 0.10] | 0.05 [0.00 to 0.09] | -0.02 [-0.05 to 0.02] | -0.01 [-0.10 to 0.08] | 0.03 [-0.03 to 0.08]
  Cycle 18 Day 1 | 0.02 [-0.06 to 0.09] | 0.01 [-0.04 to 0.07] | 0.06 [0.02 to 0.11] | -0.02 [-0.06 to 0.03] | -0.18 [-0.30 to -0.06] | 0.05 [-0.01 to 0.10]
  Cycle 20 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 20 Day 1 | -0.06 [-0.15 to 0.03] | 0.07 [0.00 to 0.13] | 0.02 [-0.05 to 0.08] | -0.01 [-0.06 to 0.05] |  | 0.02 [-0.04 to 0.09]
  Cycle 22 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 22 Day 1 | 0.02 [-0.07 to 0.11] | 0.05 [-0.02 to 0.12] | 0.04 [-0.03 to 0.11] | -0.07 [-0.14 to 0.00] |  | 0.03 [-0.04 to 0.11]
  Cycle 24 Day 1: number analyzed (Participants) | 24 | 0 | 0 | 46 | 0 | 0
  Cycle 24 Day 1 | 0.09 [-0.03 to 0.21] |  |  | 0.01 [-0.11 to 0.13] |  |
  End of treatment | -0.03 [-0.10 to 0.05] | 0.03 [-0.05 to 0.11] | 0.03 [-0.02 to 0.07] | 0.01 [-0.04 to 0.05] | -0.03 [-0.08 to 0.02] | 0.02 [-0.05 to 0.08]

70. Secondary Outcome: Change From Baseline in Total Scores for International Shopping List Test (Cognitive Function Assessment) (Phase 2)
Description: The International Shopping List task is a measure of verbal learning and uses a well validated list learning paradigm administered using a computer. High frequencies, high imagery, concrete nouns (items from a shopping list) were read to the participant at the rate of one word every 2 seconds. Once all 12 words had been read, the participant was asked to recall as many of the words as quickly as possible. The words recalled by the participant were marked on the computer screen. When the participant could recall no more words, the same list was read again. The words recalled by the participant were recorded. This was then repeated a third time. Total number of correct responses on 3 consecutive trials at a single assessment was recorded. Lower values of least square mean change from baseline indicate performance decline. Upper limit of 95% confidence interval of -0.00 or lower indicate statistically significant decline of performance over baseline at that cycle.
Time Frame: Baseline, Day 1 of Cycles 2-5, Day 1 of every other cycle from Cycle 6, and end of treatment (up to 3 years)
Population: as for outcome 66
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 24 | 26 | 50 | 46 | 38 | 29
Units on a scale
  Cycle 2 Day 1 | -0.02 [-1.89 to 1.84] | -1.13 [-2.90 to 0.64] | 0.25 [-1.01 to 1.52] | -0.45 [-1.76 to 0.86] | 0.96 [-0.50 to 2.43] | 0.16 [-1.51 to 1.83]
  Cycle 3 Day 1 | 0.19 [-1.66 to 2.03] | -0.81 [-2.58 to 0.96] | 0.14 [-1.15 to 1.43] | -1.04 [-2.36 to 0.29] | -0.08 [-1.59 to 1.44] | -0.56 [-2.21 to 1.09]
  Cycle 4 Day 1 | 0.58 [-1.26 to 2.42] | 0.26 [-1.54 to 2.05] | 0.28 [-1.05 to 1.61] | 0.24 [-1.12 to 1.60] | 1.30 [-0.26 to 2.86] | -0.87 [-2.59 to 0.84]
  Cycle 5 Day 1 | 1.30 [-0.51 to 3.12] | -0.66 [-2.53 to 1.21] | 0.59 [-0.77 to 1.95] | -0.94 [-2.33 to 0.45] | 1.23 [-0.36 to 2.82] | 0.74 [-0.97 to 2.45]
  Cycle 6 Day 1 | 0.18 [-1.64 to 1.99] | 0.81 [-1.06 to 2.68] | 0.50 [-0.87 to 1.87] | 0.08 [-1.31 to 1.47] | 0.82 [-0.83 to 2.46] | -0.51 [-2.31 to 1.29]
  Cycle 8 Day 1 | 0.84 [-1.00 to 2.68] | 0.60 [-1.30 to 2.50] | 1.69 [0.29 to 3.08] | 0.15 [-1.27 to 1.57] | 0.44 [-1.23 to 2.11] | 1.70 [-0.11 to 3.50]
  Cycle 10 Day 1 | 0.26 [-1.68 to 2.21] | 2.59 [0.65 to 4.52] | 0.86 [-0.56 to 2.27] | 0.13 [-1.46 to 1.72] | 2.29 [0.53 to 4.05] | 0.97 [-0.99 to 2.93]
  Cycle 12 Day 1 | 2.87 [0.86 to 4.88] | 0.02 [-2.06 to 2.10] | 0.11 [-1.52 to 1.73] | 0.69 [-0.98 to 2.35] | 1.74 [-0.25 to 3.72] | 3.10 [1.06 to 5.14]
  Cycle 14 Day 1 | 1.91 [-0.71 to 4.53] | 1.46 [-0.85 to 3.78] | 2.27 [0.36 to 4.17] | 0.94 [-0.86 to 2.73] | -4.43 [-7.11 to -1.75] | 2.67 [0.09 to 5.25]
  Cycle 16 Day 1 | 4.52 [1.58 to 7.46] | 0.87 [-2.06 to 3.79] | 1.36 [-1.11 to 3.84] | 1.04 [-0.99 to 3.07] | 3.46 [-1.26 to 8.18] | 1.97 [-0.93 to 4.87]
  Cycle 18 Day 1 | 4.77 [0.82 to 8.73] | 0.66 [-2.50 to 3.81] | -0.27 [-2.89 to 2.36] | -0.52 [-2.77 to 1.73] | -0.35 [-6.90 to 6.21] | 3.13 [0.00 to 6.27]
  Cycle 20 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 20 Day 1 | -2.72 [-7.47 to 2.03] | -1.44 [-4.91 to 2.03] | 0.56 [-2.81 to 3.92] | 1.20 [-1.84 to 4.24] |  | 0.56 [-2.89 to 4.01]
  Cycle 22 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 22 Day 1 | -5.72 [-10.47 to -0.97] | -0.28 [-4.22 to 3.66] | 2.17 [-1.68 to 6.01] | -0.36 [-4.21 to 3.48] |  | 3.99 [0.07 to 7.91]
  Cycle 24 Day 1: number analyzed (Participants) | 24 | 0 | 0 | 46 | 0 | 0
  Cycle 24 Day 1 | -8.49 [-15.06 to -1.92] |  |  | -3.35 [-9.86 to 3.16] |  |
  End of treatment | 1.02 [-2.99 to 5.04] | -1.62 [-5.95 to 2.71] | 0.80 [-1.80 to 3.40] | -0.27 [-2.47 to 1.92] | 2.37 [-0.54 to 5.27] | -0.60 [-4.09 to 2.89]

71. Secondary Outcome: Change From Baseline in Total Scores for International Shopping List Test-Delayed Recall (Cognitive Function Assessment) (Phase 2)
Description: This test was performed in the same way as the International Shopping List Test, with the exception that, the delayed recall condition required the participant to recall the words from the list 15 30 minutes later without having the list read again. During the recognition condition, the qualified personnel read a shopping list item that may or may not have been on the original list and the participant had to respond either affirmatively (if the item was on the original list) or negatively (if it was not). Total number of correct responses made in remembering the word list after a delay was recorded. Lower values of least square mean change from baseline indicate performance decline. Upper limit of 95% confidence interval of -0.00 or lower indicate statistically significant decline of performance over baseline at that cycle.
Time Frame: Baseline, Day 1 of Cycles 2-5, Day 1 of every other cycle from Cycle 6, and end of treatment (up to 3 years)
Population: as for outcome 66
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2)
Number analyzed (Participants) | 24 | 26 | 50 | 46 | 38 | 29
Units on a scale
  Cycle 2 Day 1 | 0.10 [-0.85 to 1.06] | -0.84 [-1.76 to 0.08] | -0.12 [-0.77 to 0.53] | -0.59 [-1.28 to 0.09] | -0.22 [-0.96 to 0.53] | -0.25 [-1.11 to 0.62]
  Cycle 3 Day 1 | -0.33 [-1.28 to 0.62] | -1.32 [-2.24 to -0.40] | -0.14 [-0.81 to 0.52] | -0.77 [-1.46 to -0.07] | -0.87 [-1.64 to -0.10] | -0.30 [-1.15 to 0.56]
  Cycle 4 Day 1 | -0.44 [-1.38 to 0.50] | -0.91 [-1.86 to 0.03] | 0.03 [-0.66 to 0.72] | -0.25 [-0.97 to 0.47] | -0.02 [-0.82 to 0.78] | -1.06 [-1.95 to -0.18]
  Cycle 5 Day 1 | -0.35 [-1.29 to 0.59] | -0.57 [-1.54 to 0.40] | 0.02 [-0.69 to 0.73] | -0.46 [-1.20 to 0.27] | 0.09 [-0.74 to 0.92] | 0.17 [-0.72 to 1.05]
  Cycle 6 Day 1 | 0.48 [-0.46 to 1.42] | -0.38 [-1.35 to 0.59] | 0.12 [-0.59 to 0.84] | -0.22 [-0.95 to 0.52] | 0.30 [-0.55 to 1.15] | -0.28 [-1.21 to 0.66]
  Cycle 8 Day 1 | 0.56 [-0.38 to 1.50] | -0.24 [-1.23 to 0.75] | 0.02 [-0.70 to 0.74] | -0.49 [-1.24 to 0.25] | -1.08 [-1.94 to -0.22] | -0.16 [-1.10 to 0.77]
  Cycle 10 Day 1 | 0.29 [-0.74 to 1.31] | 0.80 [-0.22 to 1.82] | 0.54 [-0.20 to 1.28] | 0.23 [-0.61 to 1.08] | 0.25 [-0.67 to 1.16] | -0.00 [-1.02 to 1.02]
  Cycle 12 Day 1 | 0.90 [-0.15 to 1.95] | 0.13 [-0.95 to 1.21] | 0.22 [-0.63 to 1.07] | 0.19 [-0.70 to 1.07] | 0.60 [-0.43 to 1.64] | 0.42 [-0.64 to 1.49]
  Cycle 14 Day 1 | 0.38 [-0.99 to 1.75] | 0.06 [-1.15 to 1.27] | 1.06 [0.06 to 2.06] | 0.11 [-0.85 to 1.07] | -1.80 [-3.31 to -0.30] | 0.35 [-1.00 to 1.71]
  Cycle 16 Day 1 | 0.89 [-0.66 to 2.43] | 0.52 [-1.02 to 2.05] | 0.68 [-0.62 to 1.98] | -0.12 [-1.22 to 0.98] | 0.40 [-2.09 to 2.88] | -0.22 [-1.75 to 1.30]
  Cycle 18 Day 1 | 1.06 [-1.02 to 3.14] | 0.68 [-0.98 to 2.34] | 0.38 [-1.00 to 1.76] | -0.24 [-1.54 to 1.07] | -0.39 [-3.85 to 3.07] | -0.33 [-1.97 to 1.32]
  Cycle 20 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 20 Day 1 | -1.22 [-3.73 to 1.28] | 0.16 [-1.67 to 1.98] | -0.24 [-2.01 to 1.53] | -0.18 [-1.78 to 1.43] |  | -0.70 [-2.52 to 1.11]
  Cycle 22 Day 1: number analyzed (Participants) | 24 | 26 | 50 | 46 | 0 | 29
  Cycle 22 Day 1 | -3.22 [-5.73 to -0.72] | 0.68 [-1.40 to 2.76] | 0.80 [-1.23 to 2.83] | -0.64 [-2.67 to 1.39] |  | 0.37 [-1.70 to 2.43]
  Cycle 24 Day 1: number analyzed (Participants) | 24 | 0 | 0 | 46 | 0 | 0
  Cycle 24 Day 1 | -2.43 [-5.89 to 1.04] |  |  | -0.80 [-4.25 to 2.64] |  |
  End of treatment | -0.87 [-2.99 to 1.24] | -2.31 [-4.58 to -0.04] | 0.52 [-0.84 to 1.89] | -0.85 [-2.06 to 0.35] | -0.19 [-1.71 to 1.34] | 0.11 [-1.72 to 1.95]

72. Secondary Outcome: Number of Participants With Absolute Values and Change From Baseline in PR Interval Meeting Pre-defined Criteria (Phase 2 and DDI Substudy)
Description: PR Interval was determined by ECG measurement. PR interval had following categories: change from baseline>=25 percent, 40 to <60 milliseconds (msec), 60 to <80 msec and >=80 msec. Baseline was defined as the average of the triplicate measurements prior to the first dose of study drug.
Time Frame: From first dose of study treatment to end of treatment maximum of 7.5 years for Phase 2 and up to a maximum of 6 years approx. for DDI sub study)
Population: Safety analysis set: all enrolled participants who received at least 1 dose of PF-06463922. Here, "Overall Number of Participants Analyzed": participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- DDI Substudy: Participants with advanced ALK positive or ROS1-positive NSCLC who were treatment naïve or had any number of prior cancer therapies with or without asymptomatic CNS metastases were administered a single dose of a probe substrate alone on Day -2. Participants were given PF-06463922 100 mg orally QD starting on Cycle1 Day 1 and along with probe substrate on Day 15 Cycle 1.
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Substudy
Number analyzed (Participants) | 29 | 27 | 59 | 64 | 46 | 47 | 32
Participants
  Change from baseline: >25% | 4 | 3 | 8 | 9 | 6 | 10 | 2
  Absolute value: 40-<60 msec | 3 | 2 | 2 | 2 | 3 | 7 | 2
  Absolute value: 60-<80 msec | 0 | 1 | 2 | 4 | 1 | 1 | 0
  Absolute value: >=80 msec | 1 | 0 | 0 | 1 | 1 | 2 | 0

73. Other Pre Specified Outcome: Percentage of Participants With Overall and Intracranial Objective Response (Phase 2 and DDI Sub-study)
Description: Objective response (OR) refers to confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. Intracranial OR refers to confirmed CR or PR considering only lesions within brain. CR was defined as the disappearance of all non-lymph node target lesions (where all target lesions are recorded with a length of 0 milliliter (mm) on Target Lesions eCRF). Any pathological lymph nodes (recorded as target lesion) must have reduction in short axis to <10 mm. PR was defined as a 30 percent (%) or more decrease in sum of lesion dimensions (SLD) of target lesions, taking as reference the baseline SLD. Results presented here were based on independent central review.
Time Frame: as for outcome 72
Population: ITT analysis set was used for overall response assessment and included all enrolled participants with documented ALK or ROS1 rearrangement who received at least 1 dose of PF-06463922; participants with central nervous system (CNS) metastases in the ITT analysis set were used for intracranial response assessment. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2: Participants with advanced ROS1-positive NSCLC who were treatment naïve or had any number of prior cancer therapies with or without asymptomatic CNS metastases were given PF-06463922 100 mg orally QD on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
Arm/Group | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | Phase 2 | DDI Sub-study
Number analyzed (Participants) | 30 | 27 | 60 | 65 | 46 | 47 | 32
Percentage of participants
  Objective response | 90.0 [73.5 to 97.9] | 77.8 [57.7 to 91.4] | 56.7 [43.2 to 69.4] | 40.0 [28.0 to 52.9] | 37.0 [23.2 to 52.5] | 38.3 [24.5 to 53.6] | 40.6 [23.7 to 59.4]
  Intracranial objective response: number analyzed (Participants) | 8 | 17 | 33 | 45 | 37 | 25 | 16
  Intracranial objective response | 75.0 [34.9 to 96.8] | 58.8 [32.9 to 81.6] | 66.7 [48.2 to 82.0] | 53.3 [37.9 to 68.3] | 43.2 [27.1 to 60.5] | 56.0 [34.9 to 75.6] | 25.0 [7.3 to 52.4]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to end of treatment (maximum of 96.58 months of treatment exposure for Phase 1, maximum of 89.65 months of treatment exposure for Phase 2 and maximum of 68.69 months of treatment exposure for DDI participants)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- EXP-1 (Phase 2): Treatment-naïve participants with advanced ALK-positive NSCLC with or without asymptomatic central nervous system (CNS) metastases were given PF-06463922 100 mg orally QD on Day -7 (only participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-4 (Phase 2): Participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after 2 prior lines of ALK inhibitor therapies were given PF-06463922 100 mg orally once daily (QD) on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-5 (Phase 2): Participants with advanced ALK-positive NSCLC with or without asymptomatic CNS metastases relapsing after 3 prior lines of ALK inhibitor therapies were given PF-06463922 100 mg orally once daily (QD) on Day -7 (only for participant scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
- EXP-6 (Phase 2): Participants with advanced ROS1-positive NSCLC who were treatment naïve or had any number of prior cancer therapies with or without asymptomatic CNS metastases were given PF-06463922 100 mg orally once daily (QD) on Day -7 (only for participants scheduled for pharmacokinetic evaluation) and in 21-day cycles from Cycle 1 Day 1 until progression of disease (unless clinical benefit was still achievable), unacceptable toxicity, death or consent withdrawal.
Arm/Group | 10 mg QD (Phase 1) | 25 mg QD (Phase 1) | 50 mg QD (Phase 1) | 75 mg QD (Phase 1) | 100 mg QD (Phase 1) | 150 mg QD (Phase 1) | 200 mg QD (Phase 1) | 35 mg BID (Phase 1) | 75 mg BID (Phase 1) | 100 mg BID (Phase 1) | Japan Lead-In Cohort (LIC) | EXP-1 (Phase 2) | EXP-2 (Phase 2) | EXP-3 (Phase 2) | EXP-4 (Phase 2) | EXP-5 (Phase 2) | EXP-6 (Phase 2) | DDI Substudy
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 6/12 | 9/17 | 3/3 | 2/3 | 3/3 | 2/3 | 2/4 | 1/3 | 8/30 | 13/27 | 25/60 | 46/65 | 37/46 | 22/47 | 17/32
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 1/3 | 6/12 | 10/17 | 3/3 | 2/3 | 2/3 | 2/3 | 2/4 | 1/3 | 15/30 | 11/27 | 34/60 | 31/65 | 23/46 | 21/47 | 13/32
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 12/12 | 17/17 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 30/30 | 27/27 | 59/60 | 65/65 | 45/46 | 47/47 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 10 mg QD (Phase 1) (N=3) | 25 mg QD (Phase 1) (N=3) | 50 mg QD (Phase 1) (N=3) | 75 mg QD (Phase 1) (N=12) | 100 mg QD (Phase 1) (N=17) | 150 mg QD (Phase 1) (N=3) | 200 mg QD (Phase 1) (N=3) | 35 mg BID (Phase 1) (N=3) | 75 mg BID (Phase 1) (N=3) | 100 mg BID (Phase 1) (N=4) | Japan Lead-In Cohort (LIC) (N=3) | EXP-1 (Phase 2) (N=30) | EXP-2 (Phase 2) (N=27) | EXP-3 (Phase 2) (N=60) | EXP-4 (Phase 2) (N=65) | EXP-5 (Phase 2) (N=46) | EXP-6 (Phase 2) (N=47) | DDI Substudy (N=32)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0/6 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 7 | 8 | 6 | 6 | 5
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 1 | 0 | 1 | 0
Biloma (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 5 | 2 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0/2 | 1 | 0 | 0 | 5 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/64 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0/64 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 4 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1/3 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/3 | 0 | 0 | 0 | 0 | 0/64 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary tumour thrombotic microangiopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Brainstem compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vagus nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Assisted suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impulse-control disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Schizophreniform disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0/4 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg QD (Phase 1) (N=3) | 25 mg QD (Phase 1) (N=3) | 50 mg QD (Phase 1) (N=3) | 75 mg QD (Phase 1) (N=12) | 100 mg QD (Phase 1) (N=17) | 150 mg QD (Phase 1) (N=3) | 200 mg QD (Phase 1) (N=3) | 35 mg BID (Phase 1) (N=3) | 75 mg BID (Phase 1) (N=3) | 100 mg BID (Phase 1) (N=4) | Japan Lead-In Cohort (LIC) (N=3) | EXP-1 (Phase 2) (N=30) | EXP-2 (Phase 2) (N=27) | EXP-3 (Phase 2) (N=60) | EXP-4 (Phase 2) (N=65) | EXP-5 (Phase 2) (N=46) | EXP-6 (Phase 2) (N=47) | DDI Substudy (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 7 | 3 | 1 | 1 | 2 | 2 | 0 | 6 | 2 | 6 | 18 | 7 | 7 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 5 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 3 | 2
Ventricular dysfunction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 6 | 8 | 4 | 1 | 3
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 2 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0
Presbyopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 3 | 4 | 2 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 4 | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 7 | 3 | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 7 | 6 | 3 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 0 | 4 | 5 | 2 | 1 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 4 | 0 | 2 | 1 | 1 | 0 | 0 | 9 | 8 | 11 | 8 | 9 | 5 | 8
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 4 | 1 | 2 | 0 | 0 | 3 | 0 | 11 | 6 | 12 | 22 | 9 | 9 | 5
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 2 | 2 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 6 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 5 | 4 | 0 | 3
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 7 | 2 | 3 | 4 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (3) | 1 | 0 | 3 | 4 | 0 | 1 | 0 | 1 | 3 | 1 | 6 | 7 | 9 | 18 | 10 | 9 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 3 | 10 | 9 | 8 | 6 | 2
Asthenia (General disorders) | 1 | 0 | 2 | 4 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 6 | 4 | 12 | 7 | 8 | 3 | 8
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 7 | 7 | 6 | 4 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 5 | 5 | 2 | 1 | 0 | 1 | 3 | 0 | 9 | 6 | 4 | 14 | 7 | 10 | 4
Gait disturbance (General disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 5 | 2 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 4 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 5 | 1 | 5 | 6 | 4 | 4 | 1
Oedema peripheral (General disorders) | 3 | 1 | 1 | 4 | 10 | 3 | 1 | 0 | 2 | 3 | 1 | 13 | 15 | 33 | 25 | 16 | 25 | 14
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 6 | 2 | 3 | 2
Performance status decreased (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 7 | 5 | 3 | 4
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 10 | 6 | 12 | 10 | 4 | 7 | 3
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 3
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 3 | 4 | 6 | 0 | 3 | 1
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 3 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 7 | 0 | 3 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5 | 5 | 4 | 2 | 6 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 6 | 10 | 4 | 1 | 4
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 6 | 4 | 0 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 5 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 3 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 11 | 6 | 6 | 9 | 3 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 3 | 6 | 4 | 3 | 1 | 4
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 8 | 4 | 3 | 5
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 2 | 12 | 7 | 8 | 7/7 | 1
Amino acid level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 2 | 0 | 0 | 1 | 5 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 2 | 7 | 8 | 5 | 10 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 3 | 4 | 0 | 2 | 0 | 0 | 2 | 1 | 8 | 2 | 13 | 8 | 9 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 3 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 6 | 4 | 1 | 0 | 0 | 0 | 1 | 3 | 11 | 13 | 19 | 19 | 16 | 19 | 17
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 2 | 1 | 6 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 6 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 4 | 3 | 3 | 4
Candida test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 3 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 4 | 9 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0 | 3 | 5 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 4 | 5 | 10 | 7 | 9 | 2
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 3 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 1 | 4 | 4 | 1 | 1 | 0 | 1 | 2 | 1 | 6 | 6 | 16 | 25 | 12 | 11 | 9
Cell death (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 2 | 0 | 6 | 4 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 7 | 12 | 2 | 3 | 1 | 1 | 1 | 0 | 16 | 14 | 33 | 38 | 27 | 25 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 5 | 2 | 6 | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 5 | 7 | 1 | 2 | 0 | 1 | 1 | 3 | 23 | 16 | 37 | 45 | 32 | 25 | 23
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 4 | 3 | 4 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 4 | 4 | 2 | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 5 | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 1 | 3 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 6 | 0 | 1 | 0 | 1 | 1 | 1 | 10 | 7 | 16 | 18 | 15 | 18 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 6 | 0 | 2 | 0 | 1 | 2 | 1 | 7 | 6 | 8 | 15 | 5 | 4 | 6
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 1 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 1 | 4
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 3 | 6 | 5 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 4 | 3 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 1 | 4 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 5 | 4 | 7 | 9 | 6 | 7 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 0 | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 6 | 10 | 11 | 7 | 8 | 8 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 7 | 8 | 2 | 3 | 1
Aphasia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 2 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 2
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradykinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 1 | 1 | 2 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 6 | 6 | 3 | 4 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 3 | 4 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 8 | 4 | 6 | 12 | 8 | 13 | 6
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 4 | 2 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 5 | 2 | 1 | 3
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Formication (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 4 | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 6 | 8 | 14 | 12 | 13 | 4 | 4
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 6 | 12 | 3 | 9 | 3
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 4 | 3 | 1 | 2 | 0 | 2 | 0 | 0 | 7 | 5 | 8 | 11 | 6 | 5 | 3
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 1 | 4 | 0 | 1 | 2 | 1 | 2 | 0 | 5 | 4 | 13 | 8 | 7 | 7 | 8
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 7 | 4 | 5 | 3 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep deficit (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Slow speech (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 7 | 2 | 6 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 4 | 2 | 2 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 10 | 5 | 4 | 4 | 3
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 2 | 6 | 1 | 2
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reading disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/46 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 3 | 2 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4 | 1 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 12 | 9 | 14 | 13 | 10 | 10 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 4 | 3 | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 4 | 0 | 0 | 3 | 1 | 2 | 1 | 8 | 6 | 22 | 18 | 11 | 17 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 6 | 3 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 4 | 4 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 5 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5 | 2 | 0 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 6 | 1 | 6 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 5 | 4 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 3 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 3 | 3 | 4 | 3 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 2 | 2 | 1 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 5 | 3 | 4 | 1
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 3 | 9 | 3 | 5 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 2 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/50 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 3 | 3 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 7 | 4 | 4 | 11 | 4 | 5 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 4 | 0 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 4 | 1 | 3 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 4 | 4 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1 | 3 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 3 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2
Fine motor skill dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 8 | 1 | 1 | 2 | 2
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 0 | 1 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 3 | 1 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 1 | 1 | 2 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 2 | 2 | 1 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 0 | 2 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT01970865/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT01970865/SAP_003.pdf